Once-Daily Single-Inhaler Triple versus Dual Therapy in Patients with COPD (IMPACT Trial)

**DUPLICATE IMPACT** 

May 14, 2021

NCT02164513

#### 1. RCT Details

This section provides a high-level overview of a **published** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Once-Daily Single-Inhaler Triple versus Dual Therapy in Patients with COPD (IMPACT Trial)

#### 1.2 Intended aim(s)

To assess the effect of once-daily combination of fluticasone furoate at a dose of 100 ug, umeclidinium at a dose of 62.5 ug, and vilanterol at a dose of 25 ug ("triple therapy") versus fluticasone furoate-vilanterol—at doses of 100 ug and 25 ug, respectively—on the annual rate of moderate or severe COPD exacerbations. (Note: RCT compares additional arm of umeclidinium-vilanterol).

#### 1.3 Primary endpoint for replication

The primary endpoint is the rate of moderate or severe COPD exacerbations defined as an exacerbation leading to treatment with antibiotics or systemic glucocorticoids or one resulting in hospitalization or death.

#### 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

This trial is a superiority trial. Assuming that the annual rate of moderate or severe exacerbation would be 0.80 among patients treated with triple therapy and 0.91 among those treated with fluticasone furoate-vilanterol, it was determined that approximately 4000 patients would be needed in the triple-therapy group and 4000 in the fluticasone furoate-vilanterol group to achieve 90% power to conclude superiority of triple therapy over fluticasone furoate-vilanterol at two sided alpha of 0.01.

#### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

Pneumonia (Hazard ratio, HR=1.02; 95% CI, 0.87-1.19) comparing fluticasone furoate-umeclidinium-vilanterol vs. fluticasone furoate-vilanterol.

#### 1.6 <u>Trial estimate</u>

Rate ratio, RR=0.85 (95% CI, 0.80-0.90) comparing fluticasone furoate-umeclidinium-vilanterol vs. fluticasone furoate-vilanterol during 52 weeks (Lipson et al., 2018).

#### 2. Person responsible for implementation of replication in Aetion

Hemin Lee, MD, MPH, implemented the study design in the Aetion Evidence Platform. She is not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

#### 3. Data Source(s)

Optum CDM, IBM® MarketScan®

#### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

# **Design Diagram – IMPACT TRIAL REPLICATION Cohort Entry Date (Day 0)** [Dispensation of Trelegy ellipta OR Breo ellipta] **Washout Window** (No Triple Therapy or Dual Therapy) Days [180, -1] **Enrollment assessment window** Days [180, 0] <u>INCL</u>: Age ≥ 40 Days [0] INCL: Clinical history of COPD Days [-All Data, 0] **INCL**: Use of COPD maintenance medications Days [-90,0] **INCL**: History of at least 1 COPD exacerbation Days [-365, -1] **EXCL:** Pregnancy; Alpha-1-antitrypsin deficiency Days [-180, 0] **EXCL**: Active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, pulmonary hypertension, interstitial lung disease, lung fibrosis, ARDS, other pulmonary disease Days [-90,0] **EXCL**: Lung volume reduction surgery Days [-365, 0] EXCL: HIV; SLE; Parkinson's disease; Myasthenia gravis; ACS/Unstable angina; Acute MI; Unstable liver disease Days [-180, 0] **EXCL**: Pneumonia and/or **COPD** exacerbation Days [-14,0] **EXCL**: Acute upper/lower respiratory infections Days [-7,0] **EXCL**: Electrical cardioversion; Catheter ablation; Permanent pacemaker; ICD Days [-90,0] **EXCL:** NYHA Class IV Heart Failure Days [-180, 0] EXCL: Oxygen Therapy Days [-180, 0] **EXCL:** Pulmonary rehabilitation Days [-180, 0] EXCL: Drug/alcohol abuse Days [-180, 0] **EXCL:** Long term antibiotic use Days [-180, 0] **PRIMARY OUTCOME:** <u>EXCL</u>: Use of systemic, oral, or parenteral corticosteroid Moderate or severe COPD exacerbations during treatment Days [-30,0] **Covariate Assessment Window** Days [-180, 0] **Follow Up Window** Days [1, censor<sup>a</sup>]

<sup>a</sup> Censoring criteria:

Occurrence of outcome

- Disenrollment
- Specific date reached
- Death
- Nursing home admissionEnd of index exposure

Day 0

Time

#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing triple therapy to fluticasone furoate-vilanterol users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of triple therapy or fluticasone furoate-vilanterol (index date). We will restrict the analyses to patients with a diagnosis of COPD who have been receiving daily maintenance therapy for at least 3 months prior to index date.

#### 5.2 <u>Important steps for cohort formation</u>

New use of fluticasone furoate-umeclidinium-vilanterol (exposure), and fluticasone furoate-vilanterol (comparator) is defined as no use of either therapy in 180 days prior to index date

#### 5.2.1 Eligible cohort entry dates

Market availability of fluticasone furoate-umeclidinium-vilanterol in the U.S. for management of COPD was approved by FDA on September 18, 2017

- IBM® MarketScan®: September 18, 2017 December 31, 2018 (end of available data)
- Optum CDM: September 18, 2017 June 30, 2020 (end of available data)

# 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

#### 5.3 Flowchart of the study cohort assembly

For fluticasone furoate-umeclidinium-vilanterol (triple therapy) vs. fluticasone furoate-vilanterol

| FLOWCHART | | | | |
|---|---|---|---|---|
| | Opt | tum | Marke | etscan |
| Less Excluded Patients | Remaining<br>Patients | | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78,202,636 | | 200,203,908 |

| Did not meet cohort entry criteria | -<br>77,961,768 | 240,868 | 200,099,629 | 104,279 |
|---|---|---|---|---|
| Excluded due to insufficient enrollment | -36,776 | 204,092 | -9,826 | 94,453 |
| Excluded due to prior use of referent | -91,082 | 113,010 | -57,156 | 37,297 |
| Excluded due to prior use of exposure | -25,673 | 87,337 | -3,129 | 34,168 |
| Excluded because patient qualified in >1 exposure category | -10 | 87,327 | -2 | 34,166 |
| Excluded based on Age : Exclude missing | -1 | 87,326 | 0 | 34,166 |
| Excluded based on Gender: Exclude missing | -3 | 87,323 | 0 | 34,166 |
| Excluded based on INCLUSION: Age >=40 | -5,749 | 81,574 | -6,431 | 27,735 |
| Excluded based on INCLUSION: Established clinical history of COPD | -19,242 | 62,332 | -12,995 | 14,740 |
| Excluded based on INCLUSION: COPD Maintenance Rx previous 90 days | 0 | 62,332 | 0 | 14,740 |
| Excluded based on Exclusion 1 Pregnancy | -12 | 62,320 | -6 | 14,734 |
| Excluded based on Exclusion 3 - Alpha-1-antitrypsin deficiency | -80 | 62,240 | -35 | 14,699 |
| Excluded based on Exclusion 4 lung disease including Tb, lung ca, bronchiectasis, sarcoidosis, ILD | -5,546 | 56,694 | -1,166 | 13,533 |
| Excluded based on Exclusion 5 - Lung volume reduction surgery | 0 | 56,694 | 0 | 13,533 |
| Excluded based on Exclusion 6 - HIV/Lupus, Parkinson, MG | -473 | 56,221 | -104 | 13,429 |
| Excluded based on Exclusion 7 - Pneumonia or COPD exacerbation [-14,0] | -2,191 | 54,030 | -1,321 | 12,108 |
| Excluded based on Exclusion 8 - Acute upper or lower respiratory infections [-7,0] | -1,335 | 52,695 | -415 | 11,693 |
| Excluded based on Exclusion 11 - Liver disease | -1,625 | 51,070 | -256 | 11,437 |
| Excluded based on Excl. 12a - Life threatening cardiac disease | -850 | 50,220 | -97 | 11,340 |
| Excluded based on Excl 12b Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months | -73 | 50,147 | -37 | 11,303 |
| Excluded based on Excl. 12c - NYHA Class IV Heart failure | -639 | 49,508 | -148 | 11,155 |
| Excluded based on Excl. 16 - Oxygen therapy | -1,252 | 48,256 | -47 | 11,108 |
| Excluded based on Excl. 18 - Pulmonary rehabilitation | -77 | 48,179 | -18 | 11,090 |
| Excluded based on Excl. 19 - Drug or alcohol abuse | -402 | 47,777 | -103 | 10,987 |
| Excluded based on Excl. 24a - Use of long term antibiotics >90 days | -280 | 47,497 | -57 | 10,930 |
| Excluded based on Excl. 24b - Use of corticosteroids [-30,-0]] | -3,211 | 44,286 | -684 | 10,246 |
| Final cohort | | 44,286 | | 10,246 |

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is new initiation of fluticasone furoate-umeclidinium-vilanterol. New initiation will be defined by no use of fluticasone furoate-umeclidinium-vilanterol in the prior 180 days before treatment initiation (washout period).

#### Comparator agent:

New initiators of fluticasone furoate-vilanterol. New initiation will be defined by no use of fluticasone furoate-vilanterol in the prior 180 days before treatment initiation

#### 6.2 Preliminary Covariates:

- Age
- Gender
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date.

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix A**):

- Primary outcome: Annual rate of moderate or severe COPD exacerbations during treatment
- Control outcome of interest: Pneumonia

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the primary analysis, as it targets the relative hazard of outcomes on treatment.

The follow-up will start the day after drug initiation (i.e., cohort entry date), as described in the IMPACT, and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - O Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug plus a defined grace period (i.e., 60 days after the end of the last prescription's days' supply in main analyses).

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7. Initial Feasibility Analysis

#### Aetion report name:

For fluticasone furoate-umeclidinium-vilanterol vs. fluticasone furoate-vilanterol
Optum CDM -https://bwh-dope.aetion.com/projects/details/1614/results/67127/result/0
IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1615/results/67126/result/0

Date conducted: 03/17/2021

Complete Aetion feasibility analysis using age and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

#### 8. Initial Power Assessment

#### Aetion report name:

For fluticasone furoate-umeclidinium-vilanterol vs. fluticasone furoate-vilanterol

Optum CDM - https://bwh-dope.aetion.com/projects/details/1614/results/67129/result/0 IBM® MarketScan®- https://bwh-dope.aetion.com/projects/details/1615/results/67128/result/0

Date conducted: 03/17/2021

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, gender, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

- Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.
- Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 3/19/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

For fluticasone furoate-umeclidinium-vilanterol vs. fluticasone furoate-vilanterol

Optum CDM: https://bwh-dope.aetion.com/projects/details/1614/rwrs/67810

IBM® MarketScan®: https://bwh-dope.aetion.com/projects/details/1615/rwrs/67811

Date conducted: 03/31/2021

#### 10-A. Second Power Assessment

Date conducted: 4/14/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

#### o Pooled

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 27,512 |
| Reference | 13,756 |
| Exposed | , |
| Lxposed | 13,756 |
| Risk per 1,000 patients | 169.90 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 4674.2888 |
| Power | 0.999838206 |

o Optum CDM

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 24,142 |
| Reference | 12,071 |
| Exposed | 12,071 |
| Risk per 1,000 patients | 185.24 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 4472.06408 |
| Power | 0.999743753 |

#### o <u>IBM® MarketScan®</u>

| 3,370 |
|-------------|
| 1,685 |
| 1,685 |
| 106.86 |
| 0.85 |
| 0.05 |
| 360.1182 |
| 0.338233339 |

• Stop analyses until balance and power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 4/16/2021 |
|-------------------------|--------------|----------------|-----------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 4/30/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 10-B. Final Power Assessment after Reevaluation of Study Implementation

During a protocol review that occurred after the submission of 2<sup>nd</sup> feasibility and power analysis, the study team members agree that one inclusion criteria that was marked as "not replicable in claims" could be defined using proxy definitions. A revised cohort was created and with the updated cohort, final feasibility and power analysis was conducted. The study team members confirm that this review was performed prior to the final analysis.

#### Flowchart of the Revised Study Cohort Assembly

• Revised cohort inclusion highlighted in yellow

| | Optum | | Marketscan | |
|---|---|---|---|---|
| Less Excluded Patients | Remaining<br>Patients | | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 78,779,380 | | 200,203,908 |
| Did not meet cohort entry criteria | -<br>78,538,483 | 240,897 | 200,099,629 | 104,279 |
| Excluded due to insufficient enrollment | -36,893 | 204,004 | -9,849 | 94,430 |
| Excluded due to prior use of referent | -102,649 | 101,355 | -60,845 | 33,585 |
| Excluded due to prior use of exposure | -33,482 | 67,873 | -4,000 | 29,585 |
| Excluded because patient qualified in >1 exposure category | -10 | 67,863 | -2 | 29,583 |
| Excluded based on Age : exclude missing | -1 | 67,862 | 0 | 29,583 |
| Excluded based on Gender: exclude missing | -3 | 67,859 | 0 | 29,583 |
| Excluded based on INCLUSION: Age >=40 | -5,751 | 62,108 | -6,431 | 23,152 |
| Excluded based on INCLUSION: Established clinical history of COPD | -19,257 | 42,851 | -12,995 | 10,157 |
| Excluded based on INCLUSION: COPD Maintenance Rx previous 90 days | 0 | 42,851 | 0 | 10,157 |

| Excluded based on Inclusion: COPD exacerbation 1 year prior | <mark>-17,279</mark> | <mark>25,572</mark> | <mark>-5,381</mark> | <mark>4,776</mark> |
|---|---|---|---|---|
| Excluded based on Exclusion 1 Pregnancy | -5 | 25,567 | -1 | 4,775 |
| Excluded based on Exclusion 3 - Alpha-1-antitrypsin deficiency | -39 | 25,528 | -20 | 4,755 |
| Excluded based on Exclusion 4 lung disease including Tb, lung ca, bronchiectasis, sarcoidosis, ILD | -3,141 | 22,387 | -561 | 4,194 |
| Excluded based on Exclusion 5 - Lung volume reduction surgery | 0 | 22,387 | 0 | 4,194 |
| Excluded based on Exclusion 6 - HIV/Lupus, Parkinson, MG | -250 | 22,137 | -37 | 4,157 |
| Excluded based on Exclusion 7 - Pneumonia or COPD exacerbation [-14,-0] | -4,339 | 17,798 | -924 | 3,233 |
| Excluded based on Exclusion 8 - Acute upper or lower respiratory infections [-7,-0] | -233 | 17,565 | -87 | 3,146 |
| Excluded based on Exclusion 11 - Liver disease | -541 | 17,024 | -72 | 3,074 |
| Excluded based on Excl. 12a - Life threatening cardiac disease | -311 | 16,713 | -37 | 3,037 |
| Excluded based on Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months | -19 | 16,694 | -13 | 3,024 |
| Excluded based on Excl. 12c - NYHA Class IV Heart failure | -216 | 16,478 | -53 | 2,971 |
| Excluded based on Excl. 16 - Oxygen therapy | -626 | 15,852 | -27 | 2,944 |
| Excluded based on Excl. 18 - Pulmonary rehabilitation | -36 | 15,816 | -6 | 2,938 |
| Excluded based on Excl. 19 - Drug or alcohol abuse | -115 | 15,701 | -33 | 2,905 |
| Excluded based on Excl. 24a - Use of long term antibiotics >90 days | -111 | 15,590 | -21 | 2,884 |
| Excluded based on Excl. 24b - Use of corticosteroids [-30,0]] | -882 | 14,708 | -271 | 2,613 |
| Final cohort | | 14,708 | | 2,613 |

#### **Balance Assessment of Revised Cohort**

After review of previous feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

• Provide plot of PS distributions stratified by treatment group. Note- Please refer to **Appendix B**.

- Report covariate balance after matching.
   Note- For Table 1, please refer to Appendix B.
- Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy outcome | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| Death | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| Start of an additional exposure | 220 (2.29%) | 186 (1.94%) | 34 (0.35%) |
| End of index exposure | 4,220 (44.01%) | 2,357 (24.58%) | 1,863 (19.43%) |
| Specified date reached | 3,636 (37.92%) | 1,525 (15.91%) | 2,111 (22.02%) |
| End of patient data | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) |
| End of patient enrollment | 828 (8.64%) | 409 (4.27%) | 419 (4.37%) |
| Nursing home admission, pharmacy disenrollment | 684 (7.13%) | 317 (3.31%) | 367 (3.83%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|---|---|---|
| Patient Group Optum Marketscan | | |
| Overall Patient Population | 131 [88, 240] | 107.5 [72.5, 177] |
| Referent | 119 [88, 211.5] | 108 [86, 170] |
| Exposure | 146 [88,271] | 107 [61, 188] |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | Pooled |
|-------------------------|-----------|------------------|--------|
| Risk per 1,000 patients | 292.82 | 202.84 | 278.6 |

#### **Final Power Assessment**

Optum: https://bwh-dope.aetion.com/projects/details/1614/rwrs/69652

Marketscan: https://bwh-dope.aetion.com/projects/details/1615/rwrs/69653

Date conducted: 5/6/2021

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in above section. All other parameters in the table should be the same as in Section 8.

#### o Pooled

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 9,588 |
| Reference | 4,794 |
| Exposed | 4,794 |
| Risk per 1,000 patients | 278.60 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 2671.2168 |
| Power | 0.987449189 |

#### o Optum CDM

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 8,496 |
| Reference | 4,248 |
| Exposed | 4,248 |
| Risk per 1,000 patients | 292.82 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 2487.79872 |
| Power | 0.981829103 |

#### o <u>IBM® MarketScan®</u>

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | 1,092 |
| Reference | 546 |
| Exposed | 546 |
| Risk per 1,000 patients | 202.84 |
| Desired HR from RCT | 0.85 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 221.50128 |
| Power | 0.227214863 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Shirley Wang | Date reviewed: | 5/12/2021 |
|-------------------------|--------------|----------------|-----------|
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 11. Study Confidence and Concerns

Deadline for voting on study confidence and listing concerns:

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

#### 12. Register study protocol on clinicalTrials.gov

#### **Date conducted:**

• Register the study on clinicalTrials.gov and upload this document.

#### 13. Comparative Analyses

Aetion report name:

Date conducted:

- **a.** For primary analysis:
- **b.** For sensitivity analyses:

#### 14. Requested Results

a. Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | After adjustment | | | |
|---|---|---|---|---|---|
| | Referent Exposure Std. diff. R | Referent | Exposure | Std. diff. | |
| Number of patients | | - | | | - |
| Age categories | | | | | |

#### b. Table 2: Follow-up time

| Patient Group | ient Group Median Follow-Up Time (Days) [IQR] |
|---|---|
| Overall Patient Population | |
| Referent | |
| Exposure | |

#### c. Table 3: Censoring events

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

### d. Table 4: Results from primary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; Cl, Confidence Interval.

### e. <u>Table 5: Results from secondary analyses.</u>

Effectiveness research with Real World Data to support FDA's regulatory decision making

#### 15. References

Lipson DA, Barnhart F, Brealey N, Brooks J, Criner GJ, Day NC, Dransfield MT, Halpin DMG, Han MK, Jones CE, Kilbride S, Lange P, Lomas DA, Martinez FJ, Singh D, Tabberer M, Wise RA, Pascoe SJ; IMPACT Investigators. Once-Daily Single-Inhaler Triple versus Dual Therapy in Patients with COPD. N Engl J Med. 2018 May 3;378(18):1671-1680. doi: 10.1056/NEJMoa1713901. Epub 2018 Apr 18. PMID: 29668352.

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177.

| # | IMPACT trial definitions | Implementation in routine care | References | Color Coding |
|---|---|---|---|---|
| | Trial details- clinicaltrials gov NCTO | 2164513 | Please see the following Google Drive for further details or any missing information: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-YCcnb6b-gV?usp=sharing | Criteria |
| | EXPOSURE vs. COMPARISON | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be available in the above Google Drive Folder (lisk above). ICD-9 to ICD-10 code conversions were completed using a SAS macro that implements forward/ backward mapping based on the CMS ICD-9 to ICD-10 mapping: https://www.nbcr.org/data/icd9-icd-10-cm-and-pcs-crosswalk-general-equivalence-mapping.html | Adequate mapping in claims |
| | Triple Therapy (100 μg fluticasone furoate, 62.5 μg umeclidinium [LAMA], 25 μg vilanterol [LABA]) vs. Dual Therapy (100 μg fluticasone furoate, 25 μg vilanterol [LABA] OR 62.5 μg umeclidinium [LAMA], 25 μg vilanterol [LABA]) | Exposure 100 μg fluticasone furoate, 62.5 μg umeclidinium, 25 μg vilanterol (Trelegy ellipta) Referent 100 μg fluticasone furoate, 25 μg vilanterol 6 (Breo ellipta) | | Intermediate mapping in claims |
| | PRIMARY OUTCOME | | | Poor mapping or can't be measured in claims |
| | Annual rate of moderate or severe COPD exacerbations during treatment | Measured 1 day after drug initiation in primary diagnosis position and inpatient care setting: Moderate exacerbation COPD diagnosis code occuring in inpatient any position or outpatient setting accompanied by a prescription claim for systemic steroid occuring 14 days before or after the COPD diagnosis code. Severe exacerbation COPD diagnosis code occuring in inpatient primary position COPD ICD-9: 491.*, 492.*, 496.0 ICD-10: J41.*, J42.* J43.*, J44.* | Annavarapu S, Goldfarb S, Gelb M, Moretz C, Renda A, Kaila S. Development and validation of a predictive model to identify patients at risk of severe COPD exacerbations using administrative claims data. Int J Chron Obstruct Pulmon Dis. 2018;13:2121-2130. Published 2018 Jul 11. doi:10.2147/COPD.S155773 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6805625/ | |
| | | | | Can't be measured in claims but not important for the analysis |
| H- | INCLUSION CRITERIA Informed Consent: A signed and dated written informed consent prior to study participation | N/A | | 1 |
| | Age ≥ 40 | Measured on the day of drug initiation: Age >=40 | | |
| 3 | An established clinical history of COPD in accordance with the definition by the ATS/ERS | Measure any time prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: COPD ICD-9: 491.*, 492.*, 496.0 ICD-10: J41.*, J42. * J43.*, J44.* | Annavarapu S, Goldfarb S, Gelb M, Moretz C, Renda A, Kaila S. Development and validation of a predictive model to identify patients at risk of severe COPD exacerbations using administrative claims data. Int J Chron Obstruct Pulmon Dis. 2018;13:2121-2130. Published 2018 Jul 11. doi:10.2147/COPD.S155773 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6805625/ | |
| 4 | Current or former cigarette smokers with a history of cigarette smoking of 10 pack-years at screening (visit 1) [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1 | N/A | | |
| | A score of ≥10 on the COPD Assessment Test (CAT) at screening. A post-albuterol/salbutamol FEV1/FVC ratio of <0.70 at screening. | N/A<br>N/A | | |
| _ • | A post disaction salustically in EVX/TVC1atio of No.70 at safetiming. | In/o | I . | 1 |

| 7 | Receiving daily maintenance treatment for their COPD for at least 3 months prior to Screening. | Measured 90 days prior to and including day of drug initiation with at least 1 dispensing of following COPD maintenance medications: LABA indacaterol maleate, olodaterol hcl, salmeterol xinafoate, arformoterol tartrate, formoterol fumarate, terbutaline sulfate LAMA acildinium bromide, umeclidinium bromide, tiotropium bromide, glycopyrrolate LABA/LAMA tiotropium bromide/olodaterol hcl, indacaterol maleate/glycopyrrolate, glycopyrrolate/formoterol fumarate, umeclidinium bromide/vilanterol trifenatate LABA/ICS mometasone furoate/formoterol fumarate, budesonide/formoterol fumarate, fluticasone furoate/vilanterol trifenatate, fluticasone propionate/salmeterol xinafoat | |
|---|---|---|---|
| 8 | A post-bronchodilator FEV1 < 50% predicted normal and a documented history of ≥ 1 moderate or severe COPD exacerbation in the previous 12 months OR a post-bronchodilator 50% ≤FEV1 < 80% predicted normal and a documented history of ≥ 2 moderate exacerbations or a documented history of ≥1 severe COPD exacerbation (hospitalized) in the previous 12 months. | by a prescription claim for systemic steroid occuring 14 days before or after the COPD diagnosis code. Severe exacerbation. COPD diagnosis code occuring in inpatient primary position. COPD ICD-9: 491.*, 492.*, 496.0. ICD-10: J41.*, J42. * J43.*, J44.* | Annavarapu S, Goldfarb S, Gelb M, Moretz C, Renda A, Kaila S. Development and validation of a predictive model to identify patients at risk of severe COPD exacerbations using administrative claims data. Int J Chron Obstruct Pulmon Dis. 2018;13:2121-2130. Published 2018 Jul 11. doi:10.2147/COPD.S155773 https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6805625/ |
| | alanine aminotransferase (ALT) <2x upper limit of normal (ULN); alkaline phosphatase \$1.5xULN; bilirubin \$1.5xULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) | Applied in exclusion criteria (see severe liver disease) | |
| <u> </u> | EXCLUSION CRITERIA | Assessment 400 days and a sent trade along the following trade at the second trade at | |
| 1 | Pregnacy or child bearing potential without acceptable contraceptive method | Measured 180 days prior to and including day of drug initiation in any position or any care setting: See codes in 'Pregnancy' tab | |
| 2 | Asthma - subjects with prior history of asthma are eligible if they have a current diagnosis of COPD | N/A | |
| 3 | Subjects with $lpha 1$ -antitrypsin deficiency as the underlying cause of COPD | Measured 180 days prior to and including day of drug initiation in any position or any care setting: <u>Alpha-1-antitryosin deficiency</u> ICD-9: 273.4 ICD-10: E88.01 | |

| _ | | Decree of OO decree orders and including decree described as in a control of the | 1 |
|---|---|---|---|
| 4 | Subjects with active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases | Measured 90 days prior to and including day of drug initiation in any position or any care setting: Tuberculosis ICD-9: 010.x - 018.x ICD-10: A15.x - A19.x Lung cancer ICD-9: 162.2x, 162.2x, 162.3x, 162.4x, 162.5x, 162.8x, 162.9x ICD-10: C34.0x, C34.1x, C34.2x, C34.3x, C34.8x, C34.9x Bronchiectasis ICD-9: 494.x ICD-10: 147.x Sarcoidosis ICD-9: 515.x, 516.3, 516.8, 516.9, 517.1, 517.8, 518.89 Pulmonary hypertension ICD-10: 127.0, 127.20 ICD-9: 416.0 Interstitial lung disease, lung fibrosis, ARDS ICD-9: 151.x, 516.x, 517.x, 518.8x ICD-10: 184.x, J80.x Other pulmonary disease ICD-9: 117.x | |
| 5 | Subjects with lung volume reduction surgery within the 12 months prior to screening | Measured 365 days prior to and including day of drug initiation in any position or any care setting: CPT code: 32491 32672 HCPCS code: G0305 | Decker MR, Leverson GE, Jaoude WA, Maloney JD. Lung volume reduction surgery since the National Emphysema Treatment Trial: study of Society of Thoracic Surgeons Database. J Thorac Cardiovasc Surg. 2014;148(6):2651-8.e1. doi:10.1016/j.jtcvs.2014.02.005 |
| 6 | Immune suppression (e.g. HIV, Lupus) or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis) | Measured 180 days prior to and including ay of drug initiation in any position or any care setting: HIV ICD-9: 042.x Human immunodeficiency virus [HIV] disease 079.53 Human immunodeficiency virus, type 2 [HIV-2] V08 Asymptomatic human immunodeficiency virus [HIV] infection status ICD-10: 820.x Human immunodeficiency virus [HIV] disease 897.35 Human immunodeficiency virus [HIV] disease 897.35 Human immunodeficiency virus [HIV] disease 897.35 Human immunodeficiency virus [HIV] infection status SLE ICD-9: 710.0 ICD-10: M32.x Parkinson's disease ICD-9-CM: 332.x ICD-10-CM: G20, G21.xx Myasthenia gravis ICD-9: 358.0x ICD-9: 358.0x ICD-10: G70.0x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagifilozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 |

| | I | Measured 14 days prior to and inlouding day of drug initiation in any position or any care | |
|---|---|---|---|
| 7 | Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable). In addition, any subject that experiences pneumonia and/or moderate or severe COPD exacerbation during the run-in period will be excluded | Measured 14 days prior to and inlcuding day of drug initiation in any position or any care setting: Pneumonia and or COPD exacerbation Pnuemonia ICD9: 480.x, 481.x, 482.x, 483.x, 484.x, 485.x, 486.x ICD-10: J12.x, J13.x, J14.x, J15.x, J16.x, J17.x, J18.x COPD exacerbation Moderate exacerbation COPD diagnosis code occuring in inpatient or outpatient setting, any position. For outpatient COPD diagnosis, it is accompanied by a prescription claim for systemic steroid occuring 14 days before or after the COPD diagnosis code. Severe exacerbation COPD diagnosis code occuring in inpatient primary position COPD "491.0", "491.1", "491.2", "491.2", "491.21", "491.22", "491.8", "491.9", "492.0", "J41.8", "J43.1", "J43.1" | |
| 8 | Other Respiratory tract infections that have not resolved at least 7 days prior to screening | "J43.2", "J43.9", "J44.0", "J44.1", "J47.1", "J47.9" Measured 7 days prior to and including day of drug initiation in any position or any care setting: Acute upper /lower respiratory infections ICD-9: 460.x, 461.x, 462.x, 463.x, 464.x, 461 ICD-10: J00.x, J01.x, J02.x, J03.x, J04.x, J05.x, J06.x, J20.x, J21.x, J22.x | Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure<br>Hospitalization in Routine Clinical Care: A First Analysis from the<br>Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study."<br>Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 9 | Chest x-ray (posteroanterior and lateral) reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on CXR (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a chest x-ray at Screening Visit 1 (or historical radiograph or CT scan obtained within 3 months prior to screening) that will be over-read by a central vendor. | | |
| 10 | Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled | N/A | |
| 11 | Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Note: Chronic stable hepatitis B and C are acceptable if the subject otherwise meets entry criteria | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: See codes in 'Liver disease' tab | |
| 12a | Unstable or life threatening cardiac disease: subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: ACS/unstable angina ICD-9: 411.xx Acute MI ICD-9: 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care) | |
| 12b | Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months | Measured 90 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting: Electrical cardioversion CPT: 92960, 92961 Catheter ablation CPT: 93650, 93653, 93654 93655,, 93656, 93657, 93462 Permanent pacemaker CPT: 3202-33249 Implantable cardioverter-defibrillator (ICD) ICD-9: 00.51, 00.54, 37.94 - 37.98 ICD-9: 00.51, 00.54, 37.94 - 37.98 ICD-10: 02HKOKZ, 02HK3KZ, 02HK4KZ, 02HL0KZ, 02HL3KZ, 02HL4KZ, 0JH609Z, 0JH639Z, 0JH809Z, 0JH839Z CPT-4: 33220, 33223, 33230, 33231, 33240 - 33249, 33270, 93640 - 93642, | American Medical Association, Current Procedural Terminology (CPT). Professional Edition. Chicago, IL. https://www.amaassn.org/practice-<br>management/cpt-current-procedural-terminology* https://www.cms.gov/Outreach-and-Education/MedicareLearning-<br>Network-MLN/MLNProducts/AMA-Disclaimer.html |

| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position | |
|---|---|---|---|
| 1 | | | |
| | | and inpatient or outpatient care setting: | |
| | | a v P vie | |
| | | Systolic HF | |
| 120 | NYHA Class IV Heart failure | ICD-9: 428.2x | |
| 120 | With Class Wheat Clandic | ICD-10: I50.2x | |
| | | Combined Systolic/Diastolic HF | |
| | | ICD-9: 428.4x | |
| | | ICD-10: I50.4x | |
| | Abnormal and clinically significant 12-Lead ECG finding: | N/A | |
| | - AF with rapid ventricular rate >120 BPM | , and the second | |
| | - sustained or nonsustained VT | | |
| 13 | - Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been | | |
| | inserted) | | |
| | - QTCF ≥500 msec in patients with QRS <120 msec and QTCF ≥530 msec in patients with QRS ≥ 120 msec | | |
| $\vdash$ | | N/A | |
| 14 | Contraindications: A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor<br>antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle | IN/A | |
| 14 | | | |
| $\vdash$ | glaucoma, prostatic hypertrophy or bladder neck obstruction | | |
| | Cancer: Subjects with carcinoma that has not been in complete remission for at least 5 years. Subjects who have had | N/A | |
| 15 | carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded | | |
| | based on the 5 year waiting period if the subject has been considered cured by treatment | | |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position | |
| | | and inpatient or outpatient care setting: | |
| | Owner the second live of least term (LTOT) described as section as a first term (LTOT) | | |
| 16 | Oxygen therapy: Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3L/min (Oxygen use | Home oxygen use | |
| | less than or equal to 3L/min flow is not exclusionary.) | HCPCS: E0424, E0441, E0443, | |
| | | ICD-10: Z99.81 | |
| | | ICD-9: V46. 2 | |
| | Medication prior to spirometry: Subjects who are medically unable to withhold their albuterol/salbutamol for the 4- | N/A | |
| 17 | hour period required prior to spirometry testing at each study visit | | |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position | |
| | Pulmonary rehabilitation: Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program | and inpatient or outpatient care setting: | |
| 18 | within 4 weeks prior to Screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation | | https://www.modahealth.com/pdfs/med_criteria/PulmonaryRehab.pdf |
| 10 | Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not | Pulmonary rehabilitation | nttps.//www.modaneartn.com/purs/med_criteria/rumfolid/ykelidb.pul |
| | excluded | CPT/HCPCS: G0237, G0238, G0239, G0424,S9473, 94669 | |
| $\vdash$ | | Measured 180 days prior to and including day of drug initiation in any diagnosis position | |
| 1 | | | |
| | | and inpatient or outpatient care setting: | Patorno. Elisabetta et al. "Cardiovascular outcomes associated with |
| | | and inpatient or outpatient care setting: | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population |
| 19 | Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse | and inpatient or outpatient care setting: Alcohol abuse or dependence | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 |
| 19 | Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 19 | Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Drug abuse or dependence</u> | canagliflozin versus other non-gliflozin antidiabetic drugs: population |
| 19 | | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Drug abuse or dependence</u> 292.xx, 304.xx, 305.2x-305.9x, 648.3x | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Drug abuse or dependence</u> | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 19 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Drug abuse or dependence</u> 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Drug abuse or dependence</u> 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Prug abuse or dependence</u> 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation | and inpatient or outpatient care setting: <u>Alcohol abuse or dependence</u> 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x <u>Drug abuse or dependence</u> 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivatior or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivatior or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 23 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivatior or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: - Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 23 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 23 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivatior or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: - Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20 21 22 23 | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivatior or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: - Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: See codes in 'Antibiotics' tab | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20<br>21<br>22<br>23<br>24a | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study. Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study. Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials. The use of any of the following medications under the given conditions: Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term exacerbation. | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20<br>21<br>22<br>23<br>24a | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: - Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term exacerbation Use of a systemic, oral, or parenteral corticosteroid in the last 30 days (except unless treating COPD | and inpatient or outpatient care setting: Alcohol abuse or dependence 291xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 291xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: See codes in 'Antibiotics' tab Measured 30 days prior to and including day of drug initiation: | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20<br>21<br>22<br>23<br>24a | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study. Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study. Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials. The use of any of the following medications under the given conditions: Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term exacerbation. | and inpatient or outpatient care setting: Alcohol abuse or dependence 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 292.xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: See codes in 'Antibiotics' tab Measured 30 days prior to and including day of drug initiation: Cortisone, hydrocortisone, prednisone, prednisolone, methylprednisolone, triamcinolone, | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |
| 20<br>21<br>22<br>23<br>24a | Non-compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures - any infirmity, disability, or geographic location that would limit compliance for scheduled visit. Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study Affiliation with investigator site: Study investigators, sub-investigators, study coordinators, employees of a participating investigator or study site, or immediate family members of the aforementioned that is involved with this study Inability to read: Any subject who is unable to read and/or would not be able to complete study related materials The use of any of the following medications under the given conditions: - Long term antibiotic use (short term antibiotics are allowed if treating short-term acute infection or short-term exacerbation Use of a systemic, oral, or parenteral corticosteroid in the last 30 days (except unless treating COPD | and inpatient or outpatient care setting: Alcohol abuse or dependence 291xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, E860.0x, V11.3x Drug abuse or dependence 291xx, 304.xx, 305.2x-305.9x, 648.3x N/A N/A N/A N/A N/A Measured 180 days prior to and including day of drug initiation, with days supply exceeding >90 days: See codes in 'Antibiotics' tab Measured 30 days prior to and including day of drug initiation: | canagliflozin versus other non-gliflozin antidiabetic drugs: population<br>based cohort study." BMJ 2018;360:k119 |

| Pregnancy |
|---|
| Diagnosis codes |
| 650 NORMAL DELIVERY |
| 660 OBSTRUCTED LABOR |
| 661 ABNORMALITY OF FORCES OF LABOR |
| 662 LONG LABOR |
| 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY |
| 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY |
| 665 OTHER OBSTETRICAL TRAUMA |
| 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE |
| 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND |
| DELIVERY |
| 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR |
| COMPLICATION |
| V24 POSTPARTUM CARE AND EXAMINATION |
| V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY |
| V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER |
| V24.2 ROUTINE POSTPARTUM FOLLOW |
| V27 OUTCOME OF DELIVERY |
| V27.0 MOTHER WITH SINGLE LIVEBORN |
| V27.1 MOTHER WITH SINGLE STILLBORN+A2:J81 |
| V27.2 MOTHER WITH TWINS BOTH LIVEBORN |
| V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN |
| V27.4 MOTHER WITH TWINS BOTH STILLBORN |
| V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN |
| V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN |
| V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN |
| V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY |

| D | r۸ | CO | h | | re | r | hn | ۵۵ |
|---|----|----|---|---|----|---|----|----|
| _ | u | ᇆ | u | u | | _ | - | _3 |

- 72.0 LOW FORCEPS OPERATION
- 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY
- 72.2 MID FORCEPS OPERATION
- 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY
- 72.29 OTHER MID FORCEPS OPERATION
- 72.3 HIGH FORCEPS OPERATION
- 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY
- 72.39 OTHER HIGH FORCEPS OPERATION
- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR

- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION

# **Liver Disease** 070.0 - VIRAL HEPATITIS A WITH HEPATIC COMA 070.2 - VIRAL HEPATITIS B WITH HEPATIC COMA 070.22 - CHRONIC VIRAL HEPATITIS B WITH HEPATIC COMA WITHOUT HEPATITIS DELTA 070.23 - CHRONIC VIRAL HEPATITIS B WITH HEPATIC COMA WITH HEPATITIS DELTA 070.3 - VIRAL HEPATITIS B WITHOUT MENTION OF HEPATIC COMA 070.30 - VIRAL HEPATITIS B WITHOUT HEPATIC COMA ACUTE OR UNSPECIFIED WITHOUT HEPATITIS DELTA 070.31 - VIRAL HEPATITIS B WITHOUT HEPATIC COMA ACUTE OR UNSPECIFIED WITH HEPATITIS DELTA 070.32 - CHRONIC VIRAL HEPATITIS B WITHOUT HEPATIC COMA WITHOUT HEPATITIS DELTA 070.41 - ACUTE HEPATITIS C WITH HEPATIC COMA 070.43 - HEPATITIS E WITH HEPATIC COMA 070.44 - CHRONIC HEPATITIS C WITH HEPATIC COMA 070.49 - OTHER SPECIFIED VIRAL HEPATITIS WITH HEPATIC COMA 070.51 - ACUTE HEPATITIS C WITHOUT MENTION OF HEPATIC COMA 070.54 - CHRONIC HEPATITIS C WITHOUT HEPATIC COMA 070.6 - UNSPECIFIED VIRAL HEPATITIS WITH HEPATIC COMA 070.7 - UNSPECIFIED VIRAL HEPATITIS C. 070.70 - UNSPECIFIED VIRAL HEPATITIS C WITHOUT HEPATIC COMA 070.71 - UNSPECIFIED VIRAL HEPATITIS C WITH HEPATIC COMA 456.1 - ESOPHAGEAL VARICES WITHOUT BLEEDING 456.2 - ESOPHAGEAL VARICES IN DISEASES CLASSIFIED ELSEWHERE 570 - ACUTE AND SUBACUTE NECROSIS OF LIVER 571.0 - ALCOHOLIC FATTY LIVER 571.1 - ACUTE ALCOHOLIC HEPATITIS 571.3 - ALCOHOLIC LIVER DAMAGE UNSPECIFIED 571.40 - CHRONIC HEPATITIS UNSPECIFIED 571.41 - CHRONIC PERSISTENT HEPATITIS 571.49 - OTHER CHRONIC HEPATITIS 571.5 - CIRRHOSIS OF LIVER WITHOUT ALCOHOL 571.6 - BILIARY CIRRHOSIS 571.9 - UNSPECIFIED CHRONIC LIVER DISEASE WITHOUT ALCOHOL 572.0 - ABSCESS OF LIVER





456.20 - ESOPHAGEAL VARICES IN DISEASES CLASSIFIED ELSEWHERE WITH BLEEDING 456.21 - ESOPHAGEAL VARICES IN DISEASES CLASSIFIED ELSEWHERE WITHOUT BLEEDING 571.2 - ALCOHOLIC CIRRHOSIS OF LIVER 571.4 - CHRONIC HEPATITIS 571.42 - AUTOIMMUNE HEPATITIS 571.8 - OTHER CHRONIC NONALCOHOLIC LIVER DISEASE 572.1 - PORTAL PYEMIA 572.4 - HEPATORENAL SYNDROME 573.0 - CHRONIC PASSIVE CONGESTION OF LIVER 573.2 - HEPATITIS IN OTHER INFECTIOUS DISEASES CLASSIFIED ELSEWHERE 573.3 - HEPATITIS UNSPECIFIED 573.4 - HEPATIC INFARCTION 573.5 - HEPATOPULMONARY SYNDROME 576.8 - OTHER SPECIFIED DISORDERS OF BILIARY TRACT 782.4 - JAUNDICE UNSPECIFIED NOT OF NEWBORN 789.5 - ASCITES 789.59 - OTHER ASCITES B15.9 B16.1 B16.2 B16.9 B17.0 B17.2 B17.8 B18.0 B18.1 B18.8 B19.0 B19.10 B19.21 B19.9 185.01

| • | |
|--------|---|
| 185.11 | I |
| K70.0 | |
| K70.1 | |
| K70.4 | |
| K71.2 | |
| K71.4 | ı |
| K71.5 | |
| K71.6 | |
| K71.7 | |
| K72.0 | |
| K72.1 | |
| K72.9 | |
| K72.9 | |
| K73.0 | |
| K73.2 | |
| K73.8 | |
| K74.0 | |
| K74.1 | |
| K74.2 | ı |
| K75.1 | ı |
| K75.2 | ı |
| K75.3 | |
| K75.4 | ı |
| K75.8 | |
| K75.9 | ı |
| K76.0 | ı |
| K76.1 | ı |
| K76.3 | |
| K76.5 | ı |
| K76.6 | ı |
| K76.7 | ı |
| K83.8 | |

K87 R18.0

CARBENICILLIN INDANYL SODIUM

**CEFACLOR** 

# **Antibiotics** ALATROFLOXACIN MESYLATE **AMIKACIN** AMIKACIN SULFATE AMIKACIN SULFATE IN 0.9 % SODIUM CHLORIDE AMIKACIN SULFATE/PF **AMOXICILLIN** AMOXICILLIN/POTASSIUM CLAVULANATE AMPICILLIN ANHYDROUS AMPICILLIN SODIUM AMPICILLIN SODIUM/SULBACTAM SODIUM AMPICILLIN TRIHYDRATE **AZITHROMYCIN** AZITHROMYCIN HYDROGEN CITRATE AZTREONAM AZTREONAM LYSINE AZTREONAM/DEXTROSE-WATER **BACAMPICILLIN HCL BACITRACIN BACITRACIN ZINC** BACITRACIN ZINC MICRONIZED BACITRACIN ZINC/POLYMYXIN B SULFATE BACITRACIN ZINC/POLYMYXIN B SULFATE/PRAMOXINE BACITRACIN, MICRONIZED BACITRACIN/DIMETHICONE/ZINC OXIDE **BACITRACIN/LIDOCAINE** BACITRACIN/POLYMYXIN B SULFATE BACITRACIN/POLYMYXIN B SULFATE/LIDOCAINE BACITRACIN/PRAMOXINE HCL/ALOE VERA BISMUTH SUBSALICYLATE/METRONIDAZOLE/TETRACYCLINE HCL

| T PP TIGHT I |
|-----------------------------------------------|
| CEFADROXIL |
| CEFAMANDOLE NAFATE |
| CEFAMANDOLE NAFATE/DEXTROSE 5 % IN WATER |
| CEFAZOLIN SODIUM |
| CEFAZOLIN SODIUM IN 0.9 % SODIUM CHLORIDE |
| CEFAZOLIN SODIUM/DEXTROSE 5 % IN WATER |
| CEFAZOLIN SODIUM/DEXTROSE, ISO-OSMOTIC |
| CEFAZOLIN SODIUM/WATER FOR INJECTION, STERILI |
| CEFDINIR |
| CEFDITOREN PIVOXIL |
| CEFEPIME HCL |
| CEFEPIME HCL IN DEXTROSE 5 % IN WATER |
| CEFEPIME HCL IN ISO-OSMOTIC DEXTROSE |
| CEFIXIME |
| CEFONICID SODIUM |
| CEFOPERAZONE SODIUM |
| CEFOPERAZONE SODIUM/DEXTROSE 2.4 %-WATER |
| CEFOTAXIME SODIUM |
| CEFOTAXIME SODIUM/DEXTROSE 5 % IN WATER |
| CEFOTAXIME SODIUM/DEXTROSE, ISO-OSMOTIC |
| CEFOTETAN DISODIUM |
| CEFOTETAN DISODIUM IN ISO-OSMOTIC DEXTROSE |
| CEFOTETAN IN DEXTROSE |
| CEFOXITIN SODIUM |
| CEFOXITIN SODIUM/DEXTROSE 5 % IN WATER |
| CEFOXITIN SODIUM/DEXTROSE, ISO-OSMOTIC |
| CEFPODOXIME PROXETIL |
| CEFPROZIL |
| CEFTAROLINE FOSAMIL ACETATE |
| CEFTAZIDIME |
| CEFTAZIDIME IN DEXTROSE 5% AND WATER |
| CEFTAZIDIME IN DEXTROSE, ISO-OSMOTIC |

**CEFTAZIDIME SODIUM** 

CEFTAZIDIME SODIUM IN 0.9 % SODIUM CHLORIDE

CEFTAZIDIME SODIUM IN ISO-OSMOTIC DEXTROSE

**CEFTAZIDIME/ARGININE** 

CEFTAZIDIME/AVIBACTAM SODIUM

CEFTIBUTEN

**CEFTIZOXIME SODIUM** 

CEFTIZOXIME SODIUM/DEXTROSE, ISO-OSMOTIC

CEFTOLOZANE SULFATE/TAZOBACTAM SODIUM

**CEFTRIAXONE SODIUM** 

CEFTRIAXONE SODIUM IN ISO-OSMOTIC DEXTROSE

CEFTRIAXONE SODIUM/LIDOCAINE HCL

**CEFUROXIME AXETIL** 

**CEFUROXIME SODIUM** 

CEFUROXIME SODIUM IN 0.9 % SODIUM CHLORIDE/PF

CEFUROXIME SODIUM/DEXTROSE 5 % IN WATER

CEFUROXIME SODIUM/DEXTROSE, ISO-OSMOTIC

CEFUROXIME SODIUM/WATER FOR INJECTION, STERILE

CHLORAMPHENICOL

CHLORAMPHENICOL PALMITATE

CHLORAMPHENICOL SOD SUCCINATE

CHLORAMPHENICOL/FIBRINOLYSIN/DESOXYRIBONUCLEASE

CHLOROALLYL METHENAMINE CHLORIDE

CHLORTETRACYCLINE HCL

**CINOXACIN** 

**CIPROFLOXACIN** 

CIPROFLOXACIN HCL

CIPROFLOXACIN HCL/DEXAMETHASONE

CIPROFLOXACIN HCL/FLUOCINOLONE ACETONIDE

CIPROFLOXACIN HCL/HYDROCORTISONE

CIPROFLOXACIN LACTATE

CIPROFLOXACIN LACTATE/DEXTROSE 5 % IN WATER
CIPROFLOXACIN/CIPROFLOXACIN HCL **CLARITHROMYCIN** CLINDAMYCIN HCL CLINDAMYCIN PALMITATE HCL CLINDAMYCIN PHOSPHATE CLINDAMYCIN PHOSPHATE IN 0.9 % SODIUM CHLORIDE CLINDAMYCIN PHOSPHATE/BENZOYL PEROXIDE CLINDAMYCIN PHOSPHATE/BENZOYL PEROXIDE/EMOLLIENT COMB NO.94 CLINDAMYCIN PHOSPHATE/BENZOYL PEROXIDE/HYALURONATE SODIUM CLINDAMYCIN PHOSPHATE/BENZOYL PEROXIDE/SKIN CLEANSER NO.5 CLINDAMYCIN PHOSPHATE/DEXTROSE 5 % IN WATER CLINDAMYCIN PHOSPHATE/SKIN CLEANSER COMB NO.19 CLINDAMYCIN PHOSPHATE/TRETINOIN CLOXACILLIN SODIUM COLISTIN (AS COLISTIMETHATE SODIUM) COLISTIN SULFATE COLLOIDAL BISMUTH SUBCITRATE/METRONIDAZOLE/TETRACYCLINE HCL DALBAVANCIN HCL DAPTOMYCIN DEMECLOCYCLINE HCL DICLOXACILLIN SODIUM DIRITHROMYCIN **DORIPENEM** DOXYCYCLINE CALCIUM DOXYCYCLINE HYCLATE DOXYCYCLINE HYCLATE/EYELID CLEANSER 3/EYELID EMOLLIENT NO.1 DOXYCYCLINE HYCLATE/EYELID CLEANSER NO2/EYELID CLEANSER NO3 DOXYCYCLINE HYCLATE/SKIN CLEANSER COMBINATION NO.19 DOXYCYCLINE MONOHYDRATE DOXYCYCLINE MONOHYDRATE/BENZOYL PEROXIDE DOXYCYCLINE MONOHYDRATE/OMEGA-3 COMBINATION NO.1/EYE MASK

DOXYCYCLINE MONOHYDRATE/SALICYLIC ACID/OCTINOXATE/ZINC OXIDE

DOXYCYCLINE MONOHYDRATE/SKIN CLEANSER COMBINATION NO.9 **ENOXACIN** ERTAPENEM SODIUM **ERYTHROMYCIN BASE** ERYTHROMYCIN BASE IN ETHANOL ERYTHROMYCIN BASE/BENZOYL PEROXIDE ERYTHROMYCIN ESTOLATE ERYTHROMYCIN ETHYLSUCCINATE ERYTHROMYCIN ETHYLSUCCINATE/SULFISOXAZOLE ACETYL ERYTHROMYCIN GLUCEPTATE ERYTHROMYCIN LACTOBIONATE **ERYTHROMYCIN STEARATE** FOSFOMYCIN TROMETHAMINE **GATIFLOXACIN** GATIFLOXACIN/DEXTROSE 5 % IN WATER GATIFLOXACIN/PREDNISOLONE ACETATE GATIFLOXACIN/PREDNISOLONE ACETATE/BROMFENAC SODIUM GATIFLOXACIN/PREDNISOLONE ACETATE/NEPAFENAC **GEMIFLOXACIN MESYLATE GENTAMICIN SULFATE** GENTAMICIN SULFATE IN SODIUM CHLORIDE, ISO-OSMOTIC **GENTAMICIN SULFATE/PF** GENTAMICIN SULFATE/PREDNISOLONE ACETATE GENTAMICIN SULFATE/SODIUM CHLORIDE GENTAMICIN SULFATE/SODIUM CITRATE GREPAFLOXACIN HCL IMIPENEM/CILASTATIN SODIUM KANAMYCIN SULFATE LANSOPRAZOLE/AMOXICILLIN TRIHYDRATE/CLARITHROMYCIN LEVOFLOXACIN LEVOFLOXACIN/DEXTROSE 5 % IN WATER LINCOMYCIN HCL

**LINEZOLID** 

LINEZOLID IN 0.9 % SODIUM CHLORIDE

LINEZOLID IN DEXTROSE 5 % IN WATER

LOMEFLOXACIN HCL

LORACARBEF

**MEROPENEM** 

MEROPENEM IN 0.9 % SODIUM CHLORIDE

MEROPENEM/VABORBACTAM

**METHENAMINE** 

METHENAMINE HIPPURATE

METHENAMINE MANDELATE

METHENAMINE MANDELATE/SODIUM PHOSPHATE, MONOBASIC

METHENAMINE SULFOSALICYLATE/COAL TAR/MERCURY, AMMONIATED

METHENAMINE/BENZOIC ACID/SALICYLATE/SALICYLAMIDE

METHENAMINE/METHYLENE BLUE/BENZ AC/SALICYLATE/ATROP/HYOSCY

METHENAMINE/METHYLENE BLUE/BENZOIC ACID/SALICYLAT/HYOSCYAMIN

METHENAMINE/METHYLENE BLUE/BENZOIC/PHENYL SAL/ATROPIN/HYOSCY

METHENAMINE/METHYLENE BLUE/SALICYLATE/SODIUM PHOS/HYOSCYAMIN

METHENAMINE/METHYLENE BLUE/SALICYLATE/SODIUM/HYOSCYAMINE

METHENAMINE/METHYLENE BLUE/SOD PHOS/P.SALICYLATE/HYOSCYAMINE

METHENAMINE/SOD PHOSPH, MONOBASIC/METHYLENE BLUE/HYOSCYAMINE

METHENAMINE/SODIUM PHOSPHATE, MONOBASIC

METHENAMINE/SODIUM SALICYLATE

**METRONIDAZOLE** 

METRONIDAZOLE BENZOATE

METRONIDAZOLE HCL

METRONIDAZOLE IN SODIUM CHLORIDE

METRONIDAZOLE/SKIN CLEANSER

METRONIDAZOLE/SKIN CLEANSER COMBINATION NO.23

MEZLOCILLIN SODIUM

MINOCYCLINE HCL

MINOCYCLINE HCL MICROSPHERES

MINOCYCLINE HCL/EMOL COMB NO.16/SKIN CLNSR L4/TOP AGENT NO.3 MINOCYCLINE HCL/EYELID CLEANSER COMBINATION NO. 1 MINOCYCLINE HCL/WIPES WITH SKIN CLEANSER NO.4 MOXIFLOXACIN HCL MOXIFLOXACIN HCL IN BALANCE SALT IRRIGATION SOLUTION NO.2/PF MOXIFLOXACIN HCL IN SODIUM ACETATE AND SULFATE, WATER, ISO-OSM MOXIFLOXACIN HCL IN SODIUM CHLORIDE, ISO-OSMOTIC/PF MOXIFLOXACIN HCL/DEXAMETHASONE SOD PH IN NACL, ISO-OSMOTIC/PF MOXIFLOXACIN HCL/DEXAMETHASONE SOD PH/KETOROLAC/SOD CHL/PF MOXIFLOXACIN HCL/SODIUM CHLORIDE, ISO-OSMOTIC NAFCILLIN IN DEXTROSE, ISO-OSMOTIC NAFCILLIN SODIUM NAFCILLIN SODIUM/DEXTROSE 5 % IN WATER NEOMYCIN SULF/BACITRACIN ZINC/POLYMYXIN B SULF/PRAMOXINE HCL NEOMYCIN SULF/COLISTIN SUL/HYDROCORTISONE AC/THONZONIUM BROM **NEOMYCIN SULFATE** NEOMYCIN SULFATE/BACITRACIN ZINC/POLYMYXIN B NEOMYCIN SULFATE/BACITRACIN ZINC/POLYMYXIN B SULFATE NEOMYCIN SULFATE/BACITRACIN ZINC/POLYMYXIN B/HYDROCORTISONE NEOMYCIN SULFATE/BACITRACIN ZINC/POLYMYXIN B/LIDOCAINE HCL NEOMYCIN SULFATE/BACITRACIN/COLISTIMETHATE SODIUM NEOMYCIN SULFATE/BACITRACIN/POLYMYXIN B NEOMYCIN SULFATE/BACITRACIN/POLYMYXIN B/DIPERODON NEOMYCIN SULFATE/BACITRACIN/POLYMYXIN B/LIDOCAINE NEOMYCIN SULFATE/BACITRACIN/POLYMYXIN B/PRAMOXINE NEOMYCIN SULFATE/COLISTIN SULFATE/HYDROCORTISONE NEOMYCIN SULFATE/DEXAMETHASONE SODIUM PHOSPHATE NEOMYCIN SULFATE/FLUOCINOLONE ACETONIDE NEOMYCIN SULFATE/FLUOCINOLONE ACETONIDE/EMOLLIENT COMB NO.65 NEOMYCIN SULFATE/HYDROCORTISONE NEOMYCIN SULFATE/HYDROCORTISONE ACETATE NEOMYCIN SULFATE/POLYMYXIN B SULFATE

SILVER SULFADIAZINE

NEOMYCIN SULFATE/POLYMYXIN B SULFATE/BUFFERS/HYDROCORTISONE NEOMYCIN SULFATE/POLYMYXIN B SULFATE/GRAMICIDIN D NEOMYCIN SULFATE/POLYMYXIN B SULFATE/HYDROCORTISONE NEOMYCIN SULFATE/POLYMYXIN B SULFATE/LIDOCAINE NEOMYCIN SULFATE/POLYMYXIN B SULFATE/PRAMOXINE NEOMYCIN SULFATE/POLYMYXIN B SULFATE/PREDNISOLONE NEOMYCIN/BACITRACIN/POLYMYXIN B/HYDROCORTISONE NEOMYCIN/POLYMYXIN B SULFATE/DEXAMETHASONE **NETILMICIN SULFATE NITROFURANTOIN** NITROFURANTOIN MACROCRYSTAL NITROFURANTOIN MONOHYDRATE/MACROCRYSTALS NORFLOXACIN **OFLOXACIN** OFLOXACIN/DEXTROSE 5 % IN WATER OMEPRAZOLE/CLARITHROMYCIN/AMOXICILLIN TRIHYDRATE ORITAVANCIN DIPHOSPHATE **OXACILLIN SODIUM** OXACILLIN SODIUM IN ISO-OSMOTIC DEXTROSE OXYTETRACYCLINE OXYTETRACYCLINE HCL OXYTETRACYCLINE HCL/HYDROCORTISONE ACETATE OXYTETRACYCLINE HCL/POLYMYXIN B SULFATE OXYTETRACYCLINE HCL/SULFAMETHIZOLE/PHENAZOPYRIDINE OXYTETRACYCLINE/LIDOCAINE PIPERACILLIN AND TAZOBACTAM IN DEXTROSE, ISO-OSMOTIC PIPERACILLIN SODIUM PIPERACILLIN SODIUM/DEXTROSE 5 % IN WATER PIPERACILLIN SODIUM/TAZOBACTAM SODIUM POLYMYXIN B SULFATE/TRIMETHOPRIM QUINUPRISTIN/DALFOPRISTIN

SILVER SULFADIAZINE/FOAM BANDAGE **SPARFLOXACIN** SPECTINOMYCIN HCL STREPTOMYCIN SULFATE SUCCINYLSULFATHIAZOLE SULFADIAZINE SULFADIAZINE SODIUM SULFAMERAZINE SULFAMETHOXAZOLE SULFAMETHOXAZOLE/PHENAZOPYRIDINE HCL SULFAMETHOXAZOLE/TRIMETHOPRIM SULFANILAMIDE SULFAPYRIDINE **SULFATHIAZOLE** SULFATHIAZOLE SODIUM SULFATHIAZOLE/SULFACETAMIDE/SULFABENZAMIDE SULFATHIAZOLE/SULFACETAMIDE/SULFABENZAMIDE/UREA **TEDIZOLID PHOSPHATE** TELAVANCIN HCL **TELITHROMYCIN** TETRACYCLINE TETRACYCLINE HCL TICARCILLIN DISODIUM TICARCILLIN DISODIUM/DEXTROSE 5 % IN WATER TICARCILLIN DISODIUM/POTASSIUM CLAVULANATE TINIDAZOLE TOBRAMYCIN TOBRAMYCIN IN 0.225 % SODIUM CHLORIDE **TOBRAMYCIN SULFATE** TOBRAMYCIN SULFATE/DEXTROSE 5 % IN WATER TOBRAMYCIN SULFATE/SODIUM CHLORIDE

TOBRAMYCIN/DEXAMETHASONE

TOBRAMYCIN/LOTEPREDNOL ETABONATE

TOBRAMYCIN/NEBULIZER

TRIAMCINOLONE ACETONIDE/MOXIFLOXACIN HCL/WATER/PF

TRIMETHOPRIM

TRIMETHOPRIM, MICRONIZED

TROLEANDOMYCIN

TROVAFLOXACIN MESYLATE

VANCOMYCIN HCL

VANCOMYCIN HCL/BALANCED SALT SOLUTION NO.2/PF

VANCOMYCIN IN 0.9 % SODIUM CHLORIDE

VANCOMYCIN IN 5 % DEXTROSE IN WATER

Optum MarketScan

#### BEFORE PS MATCHING





The c-statistics for the propensity score model, pre-matching was 0.786.

The postmatching c-statistic was 0.527.

The c-statistics for the propensity score model, pre-matching was 0.829.

The postmatching c-statistic was 0.577.

#### AFTER PS MATCHING





| | | | | Unn | natched | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optur | n | | Markets | can | POOLED | | | |
| Variable | Breo ellipta (dual therapy) | Trelegy ellipta (triple therapy) | St. Diff. | Breo ellipta (dual therapy) | Trelegy ellipta (triple<br>therapy) | St. Diff. | Breo ellipta (dual therapy) | Trelegy ellipta<br>(triple therapy) | St. Diff. |
| Number of patients | 7882 | 6796 | | 1873 | 730 | | 9,755 | 7,526 | |
| Year of Cohort Entry Date | | | | | | | | | |
| 2017; n (%) | 968 (12.3%) | 3 (0.0%) | 0.050 | 489 (26.1%) | 12 (1.6%) | 0.066 | 1,457 (14.9%) | 015 (0.2%) | 0.579 |
| 2018; n (%) | 3,123 (39.6%) | 1,451 (21.4%) | 0.033 | 1,384 (73.9%) | 718 (98.4%) | -0.027 | 4,507 (46.2%) | 2,169 (28.8%) | 0.365 |
| 2019; n (%) | 2,594 (32.9%) | 3,507 (51.6%) | -0.029 | NA | NA | NA | NA | NA | NA |
| 2020; n (%) | 1,197 (15.2%) | 1,835 (27.0%) | -0.026 | NA | NA | NA | NA | NA | NA |
| Age | | | | | | | | | |
| mean (sd) | 69.65 (10.15) | 70.22 (8.91) | -0.060 | 62.95 (11.21) | 64.09 (9.74) | -0.109 | 68.36 (10.36) | 69.63 (8.99) | -0.131 |
| median [IQR] | 70.00 [63.00, 77.00] | 71.00 [64.00, 77.00] | -0.105 | 61.00 [56.00, 70.00] | 62.00 [58.00, 70.00] | -0.095 | 68.27 (10.36) | 70.13 (8.99) | -0.192 |
| Age categories | | | | | | | | | |
| 40-64; n (%) | 2,264 (28.7%) | 1,703 (25.1%) | 0.007 | 1,245 (66.5%) | 480 (65.8%) | 0.001 | 3,509 (36.0%) | 2,183 (29.0%) | 0.150 |
| 65 - 74; n (%) | 3,005 (38.1%) | 2,840 (41.8%) | -0.006 | 281 (15.0%) | 121 (16.6%) | -0.004 | 3,286 (33.7%) | 2,961 (39.3%) | -0.117 |
| >= 75; n (%) | 2,613 (33.2%) | 2,253 (33.2%) | 0.000 | 347 (18.5%) | 129 (17.7%) | 0.002 | 2,960 (30.3%) | 2,382 (31.7%) | -0.030 |
| Geographic Region | | | | | | | | | ļ |
| Northeast; n (%) | 828 (10.5%) | 611 (9.0%) | 0.005 | 383 (20.4%) | 152 (20.8%) | -0.001 | 1,211 (12.4%) | 763 (10.1%) | 0.073 |
| North Central; n (%) | NA | NA | NA | 457 (24.4%) | 155 (21.2%) | 0.007 | NA | NA NA | NA |
| South; n (%) | 4,434 (56.3%) | 3,910 (57.5%) | -0.002 | 874 (46.7%) | 368 (50.4%) | -0.005 | 5,308 (54.4%) | 4,278 (56.8%) | -0.048 |
| Midwest; n (%) | 1,480 (18.8%) | 1,260 (18.5%) | 0.001 | NA NA | NA | NA | NA | NA | NA |
| West; n (%) | 1,140 (14.5%) | 1,015 (14.9%) | -0.001 | 158 (8.4%) | 55 (7.5%) | 0.003 | 1,298 (13.3%) | 1,070 (14.2%) | -0.026 |
| Unknown/Missing; n (%) | NA | NA | NA | 1 (0.1%) | 0 (0.0%) | 0.004 | NA | NA | NA |
| General Health Related Measures | IVA | IVA | INA | 1 (0.170) | 0 (0.070) | 0.004 | NA. | INA | INA |
| Smoking; n (%) | 3,293 (41.8%) | 3,589 (52.8%) | -0.016 | 604 (32.2%) | 353 (48.4%) | -0.026 | 3,897 (39.9%) | 3,942 (52.4%) | -0.253 |
| = : : : | | | -0.010 | | | -0.026 | | | -0.233 |
| Alcohol/Drug abuse or dependence; n (%) | 474 (6.0%) | 435 (6.4%) | | 67 (3.6%) | 28 (3.8%) | | 541 (5.5%) | 463 (6.2%) | |
| Obesity or Overweight; n (%) | 2,608 (33.1%) | 1,958 (28.8%) | 0.008 | 480 (25.6%) | 188 (25.8%) | 0.000 | 3,088 (31.7%) | 2,146 (28.5%) | 0.070 |
| Obesity; n (%) | 1,952 (24.8%) | 1,386 (20.4%) | 0.009 | 384 (20.5%) | 146 (20.0%) | 0.001 | 2,336 (23.9%) | 1,532 (20.4%) | 0.084 |
| Overweight; n (%) | 806 (10.2%) | 691 (10.2%) | 0.000 | 115 (6.1%) | 50 (6.8%) | -0.003 | 921 (9.4%) | 741 (9.8%) | -0.014 |
| Cardiovascular Measures | | | | | | | | | |
| Hypertension; n (%) | 6,143 (77.9%) | 5,080 (74.7%) | 0.004 | 1,171 (62.5%) | 467 (64.0%) | -0.002 | 7,314 (75.0%) | 5,547 (73.7%) | 0.030 |
| Hyperlipidemia; n (%) | 4,034 (51.2%) | 3,358 (49.4%) | 0.003 | 753 (40.2%) | 281 (38.5%) | 0.003 | 4,787 (49.1%) | 3,639 (48.4%) | 0.014 |
| MI, angina, Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 1,926 (24.4%) | 1,758 (25.9%) | -0.003 | 306 (16.3%) | 151 (20.7%) | -0.010 | 2,232 (22.9%) | 1,909 (25.4%) | -0.058 |
| Old MI; n (%) | 320 (4.1%) | 244 (3.6%) | 0.003 | 25 (1.3%) | 9 (1.2%) | 0.001 | 345 (3.5%) | 253 (3.4%) | 0.005 |
| Acute MI; n (%) | 0 (0.0%) | 0 (0.0%) | - | 10 (0.5%) | 0 (0.0%) | 0.010 | 010 (0.1%) | 000 (0.0%) | 0.045 |
| Stable angina; n (%) | 349 (4.4%) | 310 (4.6%) | -0.001 | 58 (3.1%) | 28 (3.8%) | -0.004 | 407 (4.2%) | 338 (4.5%) | -0.015 |
| Coronary atherosclerosis and other forms of chronic ischemic heart | 1,773 (22.5%) | 1,620 (23.8%) | -0.003 | 276 (14.7%) | 139 (19.0%) | -0.010 | 2,049 (21.0%) | 1,759 (23.4%) | -0.058 |
| disease; n (%) | 1,773 (22.5%) | 1,020 (23.8%) | | 2/6 (14.7%) | 139 (19.0%) | | 2,049 (21.0%) | | |
| History of CABG or PTCA; n (%) | 498 (6.3%) | 424 (6.2%) | 0.000 | 39 (2.1%) | 19 (2.6%) | -0.003 | 537 (5.5%) | 443 (5.9%) | -0.017 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%) | 379 (4.8%) | 246 (3.6%) | 0.006 | 75 (4.0%) | 17 (2.3%) | 0.010 | 454 (4.7%) | 263 (3.5%) | 0.061 |
| Stroke (Ischemic or hemorrhagic); n (%) | 222 (2.8%) | 144 (2.1%) | 0.004 | 44 (2.3%) | 10 (1.4%) | 0.007 | 266 (2.7%) | 154 (2.0%) | 0.046 |
| TIA; n (%) | 118 (1.5%) | 85 (1.3%) | 0.002 | 36 (1.9%) | 6 (0.8%) | 0.009 | 154 (1.6%) | 091 (1.2%) | 0.034 |
| Late effects of cerebrovascular disease; n (%) | 161 (2.0%) | 76 (1.1%) | 0.007 | 19 (1.0%) | 3 (0.4%) | 0.007 | 180 (1.8%) | 079 (1.0%) | 0.068 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%) | 1,380 (17.5%) | 1,095 (16.1%) | 0.003 | 223 (11.9%) | 100 (13.7%) | -0.005 | 1,603 (16.4%) | 1,195 (15.9%) | 0.014 |
| Atrial fibrillation; n (%) | 930 (11.8%) | 748 (11.0%) | 0.002 | 140 (7.5%) | 64 (8.8%) | -0.005 | 1,070 (11.0%) | 812 (10.8%) | 0.006 |
| Other cardiac dysrhythmia; n (%) | 1,380 (17.5%) | 1,095 (16.1%) | 0.003 | 223 (11.9%) | 100 (13.7%) | -0.005 | 1,603 (16.4%) | 1,195 (15.9%) | 0.014 |
| Diabetes Related Measures | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ,, | | . , | , | | ,, | , , | |
| Diabetes with or w/o complications; n (%) | 2,383 (30.2%) | 1,688 (24.8%) | 0.010 | 393 (21.0%) | 146 (20.0%) | 0.002 | 2,776 (28.5%) | 1,834 (24.4%) | 0.093 |
| Diabetes mellitus without mention of complications; n (%) | 2,071 (26.3%) | 1,462 (21.5%) | 0.010 | 336 (17.9%) | 131 (17.9%) | 0.000 | 2,407 (24.7%) | 1,593 (21.2%) | 0.083 |
| Diabetes with specified complications; n (%) | 979 (12.4%) | 617 (9.1%) | 0.010 | 129 (6.9%) | 41 (5.6%) | 0.005 | 1,108 (11.4%) | 658 (8.7%) | 0.083 |
| Diabetes with unspecified complications; n (%) | 181 (2.3%) | 144 (2.1%) | 0.010 | 47 (2.5%) | 11 (1.5%) | 0.003 | 228 (2.3%) | 155 (2.1%) | 0.030 |
| GI Conditions | 101 (2.3/0) | 144 (2.1/0) | 0.001 | 47 (2.370) | 11 (1.370) | 0.007 | 220 (2.370) | 133 (2.170) | 0.014 |
| | 2 254 (20 60/) | 1 502 (22 40/) | 0.010 | 206 (24 40/) | 144 (10 70/) | 0.003 | 2 (47 (27 40/) | 1 726 (22 40/) | 0.003 |
| GERD; n (%) | 2,251 (28.6%) | 1,592 (23.4%) | 0.010 | 396 (21.1%) | 144 (19.7%) | 0.003 | 2,647 (27.1%) | 1,736 (23.1%) | 0.092 |
| Upper GI (Diseases of esophagus, stomach and duodenum including GERD) ; n (%) | 2,432 (30.9%) | 1,730 (25.5%) | 0.010 | 451 (24.1%) | 157 (21.5%) | 0.005 | 2,883 (29.6%) | 1,887 (25.1%) | 0.101 |
| GI bleeding; n (%) | 236 (3.0%) | 152 (2.2%) | 0.005 | 40 (2.1%) | 17 (2.3%) | -0.001 | 276 (2.8%) | 169 (2.2%) | 0.038 |
| Non-infective enteritis and colitis; n (%) | 221 (2.8%) | 157 (2.3%) | 0.003 | 46 (2.5%) | 19 (2.6%) | -0.001 | 267 (2.7%) | 176 (2.3%) | 0.026 |

| Intraoperative and postprocedural complications and disorders of | 183 (2.3%) | 116 (1.7%) | 0.004 | 30 (1.6%) | 11 (1.5%) | 0.001 | 213 (2.2%) | 127 (1.7%) | 0.036 |
|---|---|---|---|---|---|---|---|---|---|
| digestive system; n (%) | ` ' | | | | | | | . , | |
| Disorders of gallbladder, biliary tract and pancreas; n (%) | 172 (2.2%) | 145 (2.1%) | 0.001 | 32 (1.7%) | 14 (1.9%) | -0.001 | 204 (2.1%) | 159 (2.1%) | 0.000 |
| Rheumatic Conditions | | | | | | | | | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n | 303 (3.8%) | 213 (3.1%) | 0.004 | 55 (2.9%) | 21 (2.9%) | 0.000 | 358 (3.7%) | 234 (3.1%) | 0.033 |
| (%) | | | | | | | | | |
| Osteoarthrosis; n (%) | 2,153 (27.3%) | 1,467 (21.6%) | 0.012 | 319 (17.0%) | 112 (15.3%) | 0.004 | 2,472 (25.3%) | 1,579 (21.0%) | 0.102 |
| Other rheumatic disorders (including gout); n (%) | 3,412 (43.3%) | 2,656 (39.1%) | 0.007 | 600 (32.0%) | 200 (27.4%) | 0.008 | 4,012 (41.1%) | 2,856 (37.9%) | 0.065 |
| Gout and other crystal arthropathies; n (%) | 302 (3.8%) | 211 (3.1%) | 0.004 | 24 (1.3%) | 6 (0.8%) | 0.005 | 326 (3.3%) | 217 (2.9%) | 0.023 |
| Other rheumatic disorders; n (%) | 3,264 (41.4%) | 2,539 (37.4%) | 0.006 | 584 (31.2%) | 198 (27.1%) | 0.008 | 3,848 (39.4%) | 2,737 (36.4%) | 0.062 |
| Neuro Conditions | | ( 1) | | | - / | | / | / | |
| Alzheimer and other Dementia Disease ; n (%) | 514 (6.5%) | 245 (3.6%) | 0.013 | 65 (3.5%) | 8 (1.1%) | 0.016 | 579 (5.9%) | 253 (3.4%) | 0.119 |
| Seizure disorders (epilepsy); n (%) | 183 (2.3%) | 80 (1.2%) | 0.008 | 16 (0.9%) | 3 (0.4%) | 0.006 | 199 (2.0%) | 083 (1.1%) | 0.073 |
| Delirium/Psychosis; n (%) | 340 (4.3%) | 169 (2.5%) | 0.010 | 48 (2.6%) | 10 (1.4%) | 0.008 | 388 (4.0%) | 179 (2.4%) | 0.091 |
| Other Conditions | 4 5 5 5 (4 0 00/) | 4 000 (45 00) | | 257 (4.4.204) | 00 (40 50) | | 4 000 (40 00) | 4 400 (45 00() | |
| Hypothyroidism; n (%) | 1,566 (19.9%) | 1,099 (16.2%) | 0.009 | 267 (14.3%) | 99 (13.6%) | 0.002 | 1,833 (18.8%) | 1,198 (15.9%) | 0.077 |
| Chronic kidney disease stages I-III; n (%) | 1,352 (17.2%) | 1,005 (14.8%) | 0.006 | 118 (6.3%) | 46 (6.3%) | 0.000 | 1,470 (15.1%) | 1,051 (14.0%) | 0.031 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 195 (2.5%) | 131 (1.9%) | 0.004 | 24 (1.3%) | 5 (0.7%) | 0.006 | 219 (2.2%) | 136 (1.8%) | 0.029 |
| COPD; n (%) | 7,071 (89.7%) | 6,609 (97.2%) | -0.008 | 1,603 (85.6%) | 709 (97.1%) | -0.012 | 8,674 (88.9%) | 7,318 (97.2%) | -0.331 |
| Asthma; n (%) | 2,558 (32.5%) | 1,198 (17.6%) | 0.030 | 710 (37.9%) | 165 (22.6%) | 0.028 | 3,268 (33.5%) | 1,363 (18.1%) | 0.358 |
| Obstructive sleep apnea; n (%) | 1,667 (21.1%) | 1,427 (21.0%) | 0.000 | 351 (18.7%) | 164 (22.5%) | -0.008 | 2,018 (20.7%) | 1,591 (21.1%) | -0.010 |
| Syncope; n (%) | 308 (3.9%) | 172 (2.5%) | 0.008 | 49 (2.6%) | 16 (2.2%) | 0.003<br>0.006 | 357 (3.7%) | 188 (2.5%) | 0.069 |
| Falls; n (%) | 571 (7.2%) | 353 (5.2%) | 0.008 | 55 (2.9%) | 14 (1.9%) | | 626 (6.4%) | 367 (4.9%) | 0.065 |
| VTE; n (%) | 259 (3.3%) | 184 (2.7%) | 0.003 | 60 (3.2%) | 9 (1.2%) | 0.013 | 319 (3.3%) | 193 (2.6%) | 0.041 |
| Combined comorbidity score, 365 days | | | | | | | | | |
| mean (sd) | 3.34 (2.76) | 3.04 (2.53) | 0.113 | 2.17 (2.14) | 2.27 (2.07) | -0.047 | 3.12 (2.65) | 2.97 (2.49) | 0.058 |
| median [IQR] | 3.00 [1.00, 5.00] | 2.00 [1.00, 4.00] | 0.378 | 1.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | -0.475 | 2.62 (2.65) | 2.00 (2.49) | 0.241 |
| INDEX 2 - Frailty Score: Empirical Version 365 days as Categories, | | | | | | | | | |
| v3 | | | | | | | | | |
| < 0.1 non frail; n (%) | 6,185 (78.5%) | 4,989 (73.4%) | 0.006 | 1,546 (82.5%) | 534 (73.2%) | 0.011 | 7,731 (79.3%) | 5,523 (73.4%) | 0.139 |
| 0.1 - < 0.2 prefrail; n (%) | 1,316 (16.7%) | 1,598 (23.5%) | -0.015 | 246 (13.1%) | 173 (23.7%) | -0.025 | 1,562 (16.0%) | 1,771 (23.5%) | -0.189 |
| > 0.2 frail; n (%) | 381 (4.8%) | 209 (3.1%) | 0.009 | 81 (4.3%) | 23 (3.2%) | 0.006 | 462 (4.7%) | 232 (3.1%) | 0.083 |
| Medication Use | | | | | | | | | |
| Use of oral corticosteroids; n (%) | 7,177 (91.1%) | 6,374 (93.8%) | -0.003 | 1,774 (94.7%) | 700 (95.9%) | -0.001 | 8,951 (91.8%) | 7,074 (94.0%) | -0.086 |
| Use of antidepressants; n (%) | 3,422 (43.4%) | 2,840 (41.8%) | 0.002 | 755 (40.3%) | 293 (40.1%) | 0.000 | 4,177 (42.8%) | 3,133 (41.6%) | 0.024 |
| Use of anticonvulsants; n (%) | 2,188 (27.8%) | 1,560 (23.0%) | 0.010 | 383 (20.4%) | 131 (17.9%) | 0.006 | 2,571 (26.4%) | 1,691 (22.5%) | 0.091 |
| Use of beta blocker OR calcium channel blocker; n (%) | 3,181 (40.4%) | 2,654 (39.1%) | 0.002 | 583 (31.1%) | 244 (33.4%) | -0.004 | 3,764 (38.6%) | 2,898 (38.5%) | 0.002 |
| Use of PPIs; n (%) | 2,956 (37.5%) | 2,205 (32.4%) | 0.009 | 611 (32.6%) | 232 (31.8%) | 0.001 | 3,567 (36.6%) | 2,437 (32.4%) | 0.088 |
| Use of opioids; n (%) | 2,762 (35.0%) | 2,042 (30.0%) | 0.009 | 587 (31.3%) | 200 (27.4%) | 0.007 | 3,349 (34.3%) | 2,242 (29.8%) | 0.097 |
| Use of antipsychotics; n (%) | 491 (6.2%) | 339 (5.0%) | 0.005 | 75 (4.0%) | 35 (4.8%) | -0.004 | 566 (5.8%) | 374 (5.0%) | 0.035 |
| Use of anxiolytics/hypnotics; n (%) | 794 (10.1%) | 651 (9.6%) | 0.002 | 189 (10.1%) | 78 (10.7%) | -0.002 | 983 (10.1%) | 729 (9.7%) | 0.013 |
| Use of dementia meds; n (%) | 290 (3.7%) | 167 (2.5%) | 0.007 | 37 (2.0%) | 4 (0.5%) | 0.013 | 327 (3.4%) | 171 (2.3%) | 0.066 |
| Use of antiparkinsonian meds; n (%) | 401 (5.1%) | 306 (4.5%) | 0.003 | 69 (3.7%) | 26 (3.6%) | 0.001 | 470 (4.8%) | 332 (4.4%) | 0.019 |
| Use of Benzodiazepine; n (%) | 1,723 (21.9%) | 1,350 (19.9%) | 0.004 | 346 (18.5%) | 149 (20.4%) | -0.004 | 2,069 (21.2%) | 1,499 (19.9%) | 0.032 |
| All antidiabetic medications; n (%) | 1,859 (23.6%) | 1,338 (19.7%) | 0.008 | 336 (17.9%) | 140 (19.2%) | -0.003 | 2,195 (22.5%) | 1,478 (19.6%) | 0.071 |
| ACEI/ARB; n (%) | 3,720 (47.2%) | 3,158 (46.5%) | 0.001 | 785 (41.9%) | 309 (42.3%) | -0.001 | 4,505 (46.2%) | 3,467 (46.1%) | 0.002 |
| Use of Anticoagulants; n (%) | 879 (11.2%) | 684 (10.1%) | 0.003 | 150 (8.0%) | 57 (7.8%) | 0.001 | 1,029 (10.5%) | 741 (9.8%) | 0.023 |
| Use of Amiodarone; n (%) | 88 (1.1%) | 76 (1.1%) | 0.000 | 13 (0.7%) | 9 (1.2%) | -0.005 | 101 (1.0%) | 085 (1.1%) | -0.010 |
| Digoxin; n (%) | 97 (1.2%) | 75 (1.1%) | 0.001 | 16 (0.9%) | 8 (1.1%) | -0.002 | 113 (1.2%) | 083 (1.1%) | 0.009 |
| Use of Diuretics; n (%) | 3,206 (40.7%) | 2,565 (37.7%) | 0.005 | 630 (33.6%) | 268 (36.7%) | -0.005 | 3,836 (39.3%) | 2,833 (37.6%) | 0.035 |
| Use of Aspirin; n (%) | 39 (0.5%) | 38 (0.6%) | -0.001 | 45 (2.4%) | 15 (2.1%) | 0.002 | 084 (0.9%) | 053 (0.7%) | 0.022 |
| NSAIDs (NOT including aspirin); n (%) | 1,489 (18.9%) | 1,151 (16.9%) | 0.005 | 379 (20.2%) | 130 (17.8%) | 0.006 | 1,868 (19.1%) | 1,281 (17.0%) | 0.055 |
| HRT (Use of estrogens, progestins, androgens); n (%) | 283 (3.6%) | 216 (3.2%) | 0.002 | 113 (6.0%) | 42 (5.8%) | 0.001 | 396 (4.1%) | 258 (3.4%) | 0.037 |
| Use of Statins ; n (%) | 4,228 (53.6%) | 3,761 (55.3%) | -0.002 | 828 (44.2%) | 317 (43.4%) | 0.001 | 5,056 (51.8%) | 4,078 (54.2%) | -0.048 |
| Healthcare Utilization Measures | | | | | | | | | |
| Use of any drugs claims | | | | | | | | | |
| mean (sd) | 39.76 (25.49) | 38.20 (22.20) | 0.065 | 36.10 (22.86) | 39.78 (22.55) | -0.162 | 39.06 (25.01) | 38.35 (22.23) | 0.030 |
| median [IQR] | 35.00 [22.00, 52.00] | 34.00 [22.00, 50.00] | 0.042 | 32.00 [20.00, 48.00] | 36.00 [23.00, 52.00] | -0.176 | 34.42 (25.01) | 34.19 (22.23) | 0.010 |
| Number of office visits | | | | | | | | | |
| mean (sd) | 19.74 (13.91) | 18.54 (12.12) | 0.092 | 14.40 (10.08) | 14.76 (9.75) | -0.036 | 18.71 (13.26) | 18.17 (11.91) | 0.043 |
| · | | | | | | | | | |

| 1 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 17.00 [10.00, 26.00] | 16.00 [10.00, 24.00] | 0.077 | 12.00 [7.00, 19.00] | 12.50 [8.00, 19.00] | -0.050 | 16.04 (13.26) | 15.66 (11.91) | 0.030 |
| Number of ED visits | 4.44(0.04) | 4 00 (4 70) | 0.460 | 4 22 (2 22) | 0.00 (4.70) | 0.445 | 4 00 (0 07) | 4 07 (4 70) | 0.450 |
| mean (sd) | 1.41 (2.24) | 1.08 (1.78) | 0.163 | 1.23 (2.39) | 0.99 (1.73) | 0.115 | 1.38 (2.27) | 1.07 (1.78) | 0.152 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 1.00] | 0.000 | 1.00 [0.00, 2.00] | 0.00 [0.00, 1.00] | 0.479 | 1.00 (2.27) | 0.90 (1.78) | 0.049 |
| Number of hospitalizations | 0.27 (0.70) | 0.46 (0.54) | 0.465 | 4 42 (2 02) | 0.04 (2.20) | 0.007 | 0.42 (4.05) | 0.22 (0.04) | 0.446 |
| mean (sd) | 0.27 (0.79) | 0.16 (0.51) | 0.165 | 1.12 (3.93) | 0.81 (2.20) | 0.097 | 0.43 (1.86) | 0.22 (0.84) | 0.146 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (1.86) | 0.00 (0.84) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%) | 253 (3.2%) | 77 (1.1%) | 0.014 | 51 (2.7%) | 7 (1.0%) | 0.013 | 304 (3.1%) | 084 (1.1%) | 0.140 |
| Old hospitalizations (-365 to -31 days); n (%) | 2,160 (27.4%) | 1,723 (25.4%) | 0.004 | 474 (25.3%) | 196 (26.8%) | -0.003 | 2,634 (27.0%) | 1,919 (25.5%) | 0.034 |
| Number of Pulmonologist visits | 0.00 (0.64) | 0.40 (0.65) | 0.046 | 0.00 (4.20) | 4 22 (4 60) | 0.200 | 0.22 (0.02) | 0.24 (0.70) | 0.025 |
| mean (sd) | 0.09 (0.64) | 0.10 (0.65) | -0.016 | 0.80 (1.38) | 1.23 (1.60) | -0.288 | 0.23 (0.83) | 0.21 (0.79) | 0.025 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 1.00] | 1.00 [0.00, 2.00] | -0.669 | 0.00 (0.83) | 0.10 (0.79) | -0.123 |
| Pulmonologist on CED ; n (%) | 44 (0.6%) | 50 (0.7%) | -0.001 | 207 (11.1%) | 75 (10.3%) | 0.002 | 251 (2.6%) | 125 (1.7%) | 0.062 |
| Number of hospital days | 2 75 (4 2 57) | 4.05 (5.40) | | 4.40 (0.00) | 0.04 (0.00) | | 2 44 (2 55) | 4.04/4.00\ | |
| mean (sd) | 2.75 (10.57) | 1.06 (5.13) | 0.203 | 1.12 (3.93) | 0.81 (2.20) | 0.097 | 2.44 (9.66) | 1.04 (4.92) | 0.183 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.000 | 0.00 (9.66) | 0.00 (4.92) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood chemistry | 5,479 (69.5%) | 4,639 (68.3%) | 0.001 | 811 (43.3%) | 344 (47.1%) | -0.006 | 6,290 (64.5%) | 4,983 (66.2%) | -0.036 |
| test; n (%) | , , , | | | | | | | | |
| Number of HbA1C test ordered | 4.47(4.46) | 4.05 (4.42) | 0.002 | 0.66 (4.45) | 0.50 (4.45) | 0.064 | 4.07 (4.44) | 4.04 (4.46) | 0.043 |
| mean (sd) | 1.17 (1.46) | 1.05 (1.42) | 0.083 | 0.66 (1.15) | 0.59 (1.15) | 0.061 | 1.07 (1.41) | 1.01 (1.40) | 0.043 |
| median [IQR] | 1.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.694 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.000 | 0.81 (1.41) | 0.00 (1.40) | 0.577 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; | 353 (4.5%) | 266 (3.9%) | 0.003 | 88 (4.7%) | 42 (5.8%) | -0.005 | 441 (4.5%) | 308 (4.1%) | 0.020 |
| n (%) Number of Mammograms (Breast cancer screening); n (%) | 1,076 (13.7%) | 786 (11.6%) | 0.006 | 220 (11.7%) | 82 (11.2%) | 0.001 | 1 200 (12 20/) | 868 (11.5%) | 0.055 |
| 5 , | | , , | | , , | , , | | 1,296 (13.3%) | . , | |
| Number of Pap smear (Cervical cancer screening); n (%) | 216 (2.7%) | 126 (1.9%) | 0.005 | 85 (4.5%) | 24 (3.3%) | 0.006 | 301 (3.1%) | 150 (2.0%) | 0.070<br>0.020 |
| Flu vaccine; n (%) | 1,701 (21.6%) | 1,389 (20.4%) | 0.003 | 329 (17.6%) | 114 (15.6%) | 0.005 | 2,030 (20.8%) | 1,503 (20.0%) | -0.020 |
| Pneumococcal vaccine; n (%) | 2,199 (27.9%) | 1,919 (28.2%) | -0.001 | 388 (20.7%) | 143 (19.6%) | 0.002 | 2,587 (26.5%) | 2,062 (27.4%) | -0.020 |
| Copay for pharmacy cost (charges in U.S. \$) | 25 22 /24 24\ | 20.00 (22.24) | -0.150 | 10.06 (10.53) | 22 20 (22 24) | 0.151 | 24.04.(20.22) | 20 22 (22 50) | -0.171 |
| mean (sd) | 25.22 (31.21) | 30.08 (33.34) | | 19.06 (19.53) | 22.29 (23.21) | -0.151 | 24.04 (29.33) | 29.32 (32.50) | |
| | 47 70 [5 47 24 40] | 22 50 57 24 44 041 | | | 40 24 [0 46 20 20] | | | | |
| median [IQR] | 17.78 [5.47, 34.48] | 22.50 [7.34, 41.01] | -0.146 | 14.94 [6.77, 25.21] | 18.31 [9.46, 28.28] | -0.157 | 17.23 (29.33) | 22.09 (32.50) | -0.157 |
| SES 9 Proxy - Business Type | | | | | | | | | |
| SES 9 Proxy - Business Type<br>Commercial; n (%) | 1,247 (15.8%) | 894 (13.2%) | 0.007 | NA | NA | NA | NA | NA | NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) | 1,247 (15.8%)<br>6,635 (84.2%) | 894 (13.2%)<br>5,902 (86.8%) | 0.007<br>-0.003 | NA<br>NA | NA<br>NA | NA<br>NA | NA<br>NA | NA<br>NA | NA<br>NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) | 1,247 (15.8%)<br>6,635 (84.2%)<br>4,493 (57.0%) | 894 (13.2%)<br>5,902 (86.8%)<br>4,227 (62.2%) | 0.007<br>-0.003<br>-0.007 | NA<br>NA<br>1,176 (62.8%) | NA<br>NA<br>514 (70.4%) | NA<br>NA<br>-0.009 | NA<br>NA<br>5,669 (58.1%) | NA<br>NA<br>4,741 (63.0%) | NA<br>NA<br>-0.100 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) | 1,247 (15.8%)<br>6,635 (84.2%)<br>4,493 (57.0%)<br>337 (4.3%) | 894 (13.2%)<br>5,902 (86.8%)<br>4,227 (62.2%)<br>309 (4.5%) | 0.007<br>-0.003<br>-0.007<br>-0.001 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%) | NA<br>NA<br>-0.009<br>-0.008 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%) | NA<br>NA<br>-0.100<br>-0.024 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) SABA/SAMA Copy; n (%) | 1,247 (15.8%)<br>6,635 (84.2%)<br>4,493 (57.0%)<br>337 (4.3%)<br>1,282 (16.3%) | 894 (13.2%)<br>5,902 (86.8%)<br>4,227 (62.2%)<br>309 (4.5%)<br>1,384 (20.4%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%)<br>276 (14.7%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) | 1,247 (15.8%)<br>6,635 (84.2%)<br>4,493 (57.0%)<br>337 (4.3%)<br>1,282 (16.3%)<br>1,736 (22.0%) | 894 (13.2%)<br>5,902 (86.8%)<br>4,227 (62.2%)<br>309 (4.5%)<br>1,384 (20.4%)<br>1,356 (20.0%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%)<br>276 (14.7%)<br>443 (23.7%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) | 1,247 (15.8%)<br>6,635 (84.2%)<br>4,493 (57.0%)<br>337 (4.3%)<br>1,282 (16.3%)<br>1,736 (22.0%)<br>61 (0.8%) | 894 (13.2%)<br>5,902 (86.8%)<br>4,227 (62.2%)<br>309 (4.5%)<br>1,384 (20.4%)<br>1,356 (20.0%)<br>73 (1.1%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%)<br>276 (14.7%)<br>443 (23.7%)<br>17 (0.9%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%)<br>12 (1.6%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) | 1,247 (15.8%)<br>6,635 (84.2%)<br>4,493 (57.0%)<br>337 (4.3%)<br>1,282 (16.3%)<br>1,736 (22.0%)<br>61 (0.8%)<br>1,635 (20.7%) | 894 (13.2%)<br>5,902 (86.8%)<br>4,227 (62.2%)<br>309 (4.5%)<br>1,384 (20.4%)<br>1,356 (20.0%)<br>73 (1.1%)<br>1,458 (21.5%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003<br>-0.002 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%)<br>12 (1.6%)<br>228 (31.2%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031<br>-0.010 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA (Sopy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA (Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LABA/ICS Combination Copy; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003<br>-0.002<br>0.084 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%)<br>276 (14.7%)<br>443 (23.7%)<br>17 (0.9%)<br>513 (27.4%)<br>1,873 (100.0%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%)<br>12 (1.6%)<br>228 (31.2%)<br>319 (43.7%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031<br>-0.010<br>1.997 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LABA/ICS Combination Copy; n (%) LAMA/LABA Combination Copy; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003<br>-0.002<br>0.084<br>-0.040 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%)<br>276 (14.7%)<br>443 (23.7%)<br>17 (0.9%)<br>513 (27.4%)<br>1,873 (100.0%)<br>88 (4.7%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%)<br>12 (1.6%)<br>228 (31.2%)<br>319 (43.7%)<br>179 (24.5%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>0.067<br>-0.052 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%)<br>456 (4.7%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031<br>-0.010<br>1.997<br>-0.446 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SAMA; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LABA Copy; n (%) LABA LABA Combination Copy; n (%) LABA/LABA Combination Copy; n (%) LABA LAMA ICS Copy; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003<br>-0.002<br>0.084<br>-0.040<br>-0.142 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.067<br>-0.052<br>-0.142 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%)<br>456 (4.7%)<br>000 (0.0%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031<br>-0.010<br>1.997<br>-0.446 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LAMA/LABA Combination Copy; n (%) LAMA/LABA Combination Copy; n (%) GOLD C/D status; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003<br>-0.002<br>0.084<br>-0.040<br>-0.142<br>-0.014 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%)<br>456 (4.7%)<br>000 (0.0%)<br>6,177 (63.3%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031<br>-0.010<br>1.997<br>-0.446<br>- |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA (copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LAMA/LABA Combination Copy; n (%) LAMA/LABA Combination Copy; n (%) LABA LAMA ICS Copy; n (%) DABA LAMA ICS Copy; n (%) SABA (CS SABA) SABA (CS Copy; n (%) SABA (CS SABA) SABA | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>0.004<br>-0.003<br>-0.002<br>0.084<br>-0.040<br>-0.142<br>-0.014 | NA<br>NA<br>1,176 (62.8%)<br>72 (3.8%)<br>276 (14.7%)<br>443 (23.7%)<br>17 (0.9%)<br>513 (27.4%)<br>1,873 (100.0%)<br>88 (4.7%)<br>0 (0.0%)<br>1,067 (57.0%)<br>9 (0.5%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%)<br>12 (1.6%)<br>228 (31.2%)<br>319 (43.7%)<br>179 (24.5%)<br>730 (100.0%)<br>537 (73.6%)<br>3 (0.4%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021<br>-0.001 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%)<br>456 (4.7%)<br>000 (0.0%)<br>6,177 (63.3%)<br>036 (0.4%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>0.036<br>-0.031<br>-0.010<br>1.997<br>-0.446<br>-<br>-0.291<br>0.017 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA/LABA Combination Copy; n (%) LAMA/LABA Combination Copy; n (%) LABA LAMA ICS Copy; n (%) GOLD C/D status; n (%) Blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>-0.004<br>-0.003<br>-0.002<br>-0.084<br>-0.040<br>-0.142<br>-0.014<br>-0.000<br>0.005 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) | NA<br>NA<br>514 (70.4%)<br>41 (5.6%)<br>143 (19.6%)<br>206 (28.2%)<br>12 (1.6%)<br>228 (31.2%)<br>319 (43.7%)<br>179 (24.5%)<br>730 (100.0%)<br>537 (73.6%)<br>3 (0.4%)<br>19 (2.6%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021<br>-0.001 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%)<br>456 (4.7%)<br>000 (0.0%)<br>6,177 (63.3%)<br>036 (0.4%)<br>264 (2.7%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%) | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.4460.291 0.017 0.053 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) SABA/ICS Combination Copy; n (%) LABA/ICS Copy; n (%) SABA/ICS Combination Copy; n (%) LABA/ICS Copy; n (%) SABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) | 0.007<br>-0.003<br>-0.001<br>-0.010<br>-0.010<br>-0.004<br>-0.003<br>-0.002<br>-0.084<br>-0.040<br>-0.142<br>-0.014<br>0.005<br>0.005 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021<br>-0.001<br>-0.004 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%) | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.446 0.291 0.017 0.053 0.029 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) SABA/SAMA Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) GOLD C/D status; n (%) blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Oxygen codes; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>-0.004<br>-0.003<br>-0.002<br>-0.084<br>-0.040<br>-0.142<br>-0.014<br>-0.005<br>-0.005<br>-0.005<br>-0.003<br>-0.003 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021<br>-0.001<br>-0.004<br>-0.004<br>-0.004 | NA<br>NA<br>5,669 (58.1%)<br>409 (4.2%)<br>1,558 (16.0%)<br>2,179 (22.3%)<br>078 (0.8%)<br>2,148 (22.0%)<br>9,755 (100.0%)<br>456 (4.7%)<br>000 (0.0%)<br>6,177 (63.3%)<br>036 (0.4%)<br>264 (2.7%)<br>816 (8.4%)<br>719 (7.4%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%) | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.4460.291 0.017 0.053 0.029 -0.206 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/LABA Combination Copy; n (%) BABA/ICS Combination Copy; n (%) SABA/ICS Combination Copy; n (%) LABA LAMA ICS Copy; n (%) SOLD C/D status; n (%) blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) | 0.007<br>-0.003<br>-0.001<br>-0.010<br>-0.010<br>-0.004<br>-0.003<br>-0.002<br>-0.084<br>-0.040<br>-0.142<br>-0.014<br>0.005<br>0.005 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021<br>-0.001<br>-0.004 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%) | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.446 0.291 0.017 0.053 0.029 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LAMA/LABA Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA LAMA ICS Copy; n (%) GOLD C/D status; n (%) blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) Insurance Plan Type | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) | 0.007<br>-0.003<br>-0.007<br>-0.001<br>-0.010<br>-0.003<br>-0.002<br>-0.084<br>-0.040<br>-0.142<br>-0.014<br>-0.000<br>0.005<br>0.003<br>-0.015 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 43 (5.9%) 43 (5.9%) 86 (11.8%) 108 (14.8%) | NA<br>NA<br>-0.009<br>-0.008<br>-0.012<br>-0.009<br>-0.006<br>-0.007<br>-0.052<br>-0.142<br>-0.021<br>-0.001<br>-0.004<br>-0.004<br>-0.019<br>-0.017 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>-0.036<br>-0.031<br>-0.010<br>1.997<br>-0.446<br>-<br>-0.291<br>-0.017<br>0.053<br>0.029<br>-0.206<br>-0.167 |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA/LABA Combination Copy; n (%) LAMA/LABA Combination Copy; n (%) GOLD C/D status; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) Insurance Plan TypeComprehensive; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) | 0.007 -0.003 -0.001 -0.010 -0.010 -0.004 -0.003 -0.0084 -0.040 -0.142 -0.014 0.000 -0.005 0.003 -0.019 -0.015 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) | NA NA -0.009 -0.008 -0.012 -0.009 -0.006 -0.007 -0.067 -0.052 -0.142 -0.021 -0.001 -0.004 -0.019 -0.017 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>5,72 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%) | NA NA O-100 O-0.024 O-112 O-0.36 O-0.31 O-0.010 I-997 O-446 - O-291 O-0.053 O-0.29 O-206 O-1.67 NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) SET COPY; n (%) GOLD C/D status; n (%) Blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) Insurance Plan TypeComprehensive; n (%)HMO; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) NA NA | 0.007 -0.003 -0.001 -0.010 -0.010 -0.004 -0.003 -0.002 -0.0084 -0.040 -0.142 -0.014 0.0005 0.003 -0.019 -0.015 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) 190 (10.1%) 195 (10.4%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) 76 (10.4%) | NA NA -0.009 -0.008 -0.012 -0.009 -0.006 -0.007 -0.052 -0.142 -0.021 -0.004 -0.004 -0.019 -0.017 -0.010 -0.000 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) NA NA | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%) | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.4460.291 0.017 0.053 0.029 -0.206 -0.167 NA NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA, SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA LABA Combination Copy; n (%) LABA LABA Combination Copy; n (%) BOLD C/D status; n (%) BOLD C/D | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) NA NA | 0.007 -0.003 -0.007 -0.001 -0.010 -0.004 -0.002 -0.084 -0.040 -0.142 -0.014 -0.005 -0.005 -0.005 -0.019 -0.015 -0.015 -0.015 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) | NA NA S14 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) 76 (10.4%) 380 (52.1%) | NA NA -0.009 -0.008 -0.012 -0.009 -0.006 -0.007 -0.052 -0.142 -0.021 -0.004 -0.004 -0.019 -0.017 -0.010 -0.000 -0.000 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) NA NA | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%) | NA<br>NA<br>-0.100<br>-0.024<br>-0.112<br>-0.036<br>-0.036<br>-0.010<br>1.997<br>-0.446<br> |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LAMA LOS Combination Copy; n (%) LABA LICS Combination Copy; n (%) GOLD C/D status; n (%) blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Nygen codes; n (%) Respiratory arrest/ dependence on oxygen; n (%) Insurance Plan TypeComprehensive; n (%)HMO; n (%)PPO; n (%)PPO; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) NA NA | 0.007 -0.003 -0.001 -0.010 -0.010 -0.004 -0.003 -0.002 -0.0084 -0.040 -0.142 -0.014 0.0005 0.003 -0.019 -0.015 | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) 190 (10.1%) 195 (10.4%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) 76 (10.4%) | NA NA -0.009 -0.008 -0.012 -0.009 -0.006 -0.007 -0.052 -0.142 -0.021 -0.004 -0.004 -0.019 -0.017 -0.010 -0.000 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) NA NA | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%) | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.4460.291 0.017 0.053 0.029 -0.206 -0.167 NA NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LAMALABA Combination Copy; n (%) LABA LAMA ICS Copy; n (%) GOLD C/D status; n (%) blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) H2 blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) Insurance Plan TypeComprehensive; n (%)HMO; n (%)PPO; n (%)DHers; n (%) Metropolitan Statistical Area | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) NA NA NA NA | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) NA NA NA NA NA | 0.007 -0.003 -0.007 -0.001 -0.010 -0.004 -0.003 -0.002 -0.084 -0.040 -0.142 -0.014 -0.003 -0.005 -0.003 -0.019 -0.015 NA NA NA NA | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) 190 (10.1%) 195 (10.4%) 1,021 (54.5%) 467 (24.9%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) 76 (10.4%) 380 (52.1%) 176 (24.1%) | NA NA O-0.009 O-0.008 O-0.12 O-0.009 O-0.007 O-0.067 O-0.052 O-1.42 O-0.011 O-0.004 O-0.004 O-0.019 O-0.017 O-0.010 O-0.000 O-0.003 O-0.002 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) NA NA NA NA NA | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%)<br>NA<br>NA<br>NA | NA NA -0.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.4460.291 0.017 0.053 0.029 -0.206 -0.167 NA NA NA NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) COD COP STATES (%) GOLD C/D STATES; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) HZ blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) Insurance Plan TypeComprehensive; n (%)PPO; n (%)PPO; n (%)Others; n (%) Metropolitan Statistical AreaUrban; n (%) | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) NA NA NA NA | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) NA NA NA NA | 0.007 -0.003 -0.001 -0.010 -0.010 -0.004 -0.003 -0.0084 -0.040 -0.142 -0.014 0.000 0.005 0.003 -0.019 -0.015 NA NA NA NA | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) 190 (10.1%) 195 (10.4%) 1,021 (54.5%) 467 (24.9%) | NA NA 14 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) 76 (10.4%) 380 (52.1%) 176 (24.1%) | NA NA O-0.009 O-0.008 O-0.12 O-0.009 O-0.067 O-0.052 O-1.42 O-0.021 O-0.004 O-0.004 O-0.017 O-0.017 O-0.010 O-0.003 O-0.002 O-0.003 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) NA NA NA NA | NA NA 4,741 (63.0%) 350 (4.7%) 1,527 (20.3%) 1,562 (20.8%) 085 (1.1%) 1,686 (22.4%) 2,512 (33.4%) 1,407 (18.7%) 7,526 (100.0%) 5,756 (76.5%) 026 (0.3%) 144 (1.9%) 572 (7.6%) 1,031 (13.7%) 1,193 (15.9%) NA NA NA NA | NA NA O.100 O.024 O.112 O.036 O.031 O.010 I.997 O.446 - O.291 O.017 O.053 O.029 O.206 O.167 NA NA NA NA |
| SES 9 Proxy - Business TypeCommercial; n (%)Medicare; n (%) SABA Copy; n (%) SABA/SAMA Copy; n (%) ICS Copy; n (%) LABA Copy; n (%) LABA Copy; n (%) LAMA Copy; n (%) LAMA Copy; n (%) LAMALICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) LABA/ICS Combination Copy; n (%) GOLD C/D status; n (%) blood eosinophilia test; n (%) Serum immunoglobulin E (IgE) level test Copy; n (%) HZ blocker; n (%) Oxygen codes; n (%) Respiratory arrest/dependence on oxygen; n (%) Insurance Plan TypeComprehensive; n (%)HMO; n (%)PPO; n (%)Dothers; n (%) Metropolitan Statistical Area | 1,247 (15.8%) 6,635 (84.2%) 4,493 (57.0%) 337 (4.3%) 1,282 (16.3%) 1,736 (22.0%) 61 (0.8%) 1,635 (20.7%) 7,882 (100.0%) 368 (4.7%) 0 (0.0%) 5,110 (64.8%) 27 (0.3%) 204 (2.6%) 686 (8.7%) 604 (7.7%) 841 (10.7%) NA NA NA NA | 894 (13.2%) 5,902 (86.8%) 4,227 (62.2%) 309 (4.5%) 1,384 (20.4%) 1,356 (20.0%) 73 (1.1%) 1,458 (21.5%) 2,193 (32.3%) 1,228 (18.1%) 6,796 (100.0%) 5,219 (76.8%) 23 (0.3%) 125 (1.8%) 529 (7.8%) 945 (13.9%) 1,085 (16.0%) NA NA NA NA NA | 0.007 -0.003 -0.007 -0.001 -0.010 -0.004 -0.003 -0.002 -0.084 -0.040 -0.142 -0.014 -0.003 -0.005 -0.003 -0.019 -0.015 NA NA NA NA | NA NA 1,176 (62.8%) 72 (3.8%) 276 (14.7%) 443 (23.7%) 17 (0.9%) 513 (27.4%) 1,873 (100.0%) 88 (4.7%) 0 (0.0%) 1,067 (57.0%) 9 (0.5%) 60 (3.2%) 130 (6.9%) 115 (6.1%) 166 (8.9%) 190 (10.1%) 195 (10.4%) 1,021 (54.5%) 467 (24.9%) | NA NA 514 (70.4%) 41 (5.6%) 143 (19.6%) 206 (28.2%) 12 (1.6%) 228 (31.2%) 319 (43.7%) 179 (24.5%) 730 (100.0%) 537 (73.6%) 3 (0.4%) 19 (2.6%) 43 (5.9%) 86 (11.8%) 108 (14.8%) 98 (13.4%) 76 (10.4%) 380 (52.1%) 176 (24.1%) | NA NA O-0.009 O-0.008 O-0.12 O-0.009 O-0.007 O-0.067 O-0.052 O-1.42 O-0.011 O-0.004 O-0.004 O-0.019 O-0.017 O-0.010 O-0.000 O-0.003 O-0.002 | NA NA 5,669 (58.1%) 409 (4.2%) 1,558 (16.0%) 2,179 (22.3%) 078 (0.8%) 2,148 (22.0%) 9,755 (100.0%) 456 (4.7%) 000 (0.0%) 6,177 (63.3%) 036 (0.4%) 264 (2.7%) 816 (8.4%) 719 (7.4%) 1,007 (10.3%) NA NA NA NA NA | NA<br>NA<br>4,741 (63.0%)<br>350 (4.7%)<br>1,527 (20.3%)<br>1,562 (20.8%)<br>085 (1.1%)<br>1,686 (22.4%)<br>2,512 (33.4%)<br>1,407 (18.7%)<br>7,526 (100.0%)<br>5,756 (76.5%)<br>026 (0.3%)<br>144 (1.9%)<br>572 (7.6%)<br>1,031 (13.7%)<br>1,193 (15.9%)<br>NA<br>NA<br>NA | NA NA O.100 -0.024 -0.112 0.036 -0.031 -0.010 1.997 -0.4460.291 -0.206 -0.167 NA NA NA NA |

Aetion link to Optum results: https://bwh-dope.aetion.com/projects/details/1614/rwrs/69652
Aetion link to Marketscan results: https://bwh-dope.aetion.com/projects/details/1615/rwrs/69653

| | | PS-ma | | | OLED | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Optum | | | Marketscan | | | | OLED | |
| Variable | Breo ellipta (dual therapy) | Trelegy ellipta (triple<br>therapy) | St. Diff. | Breo ellipta (dual therapy) | Trelegy ellipta (triple therapy) | St. Diff. | Breo ellipta<br>(dual therapy) | Trelegy ellipta<br>(triple therapy) | St. Diff |
| Number of patients | 4248 | 4248 | | 546 | 546 | | 4,794 | 4,794 | |
| Year of Cohort Entry Date | | | | | | | | | |
| 2017; n (%) | 3 (0.1%) | 3 (0.1%) | 0.0000 | 9 (1.6%) | 12 (2.2%) | -0.0044 | 012 (0.3%) | 015 (0.3%) | 0.000 |
| 2018; n (%) | 1,216 (28.6%) | 1,236 (29.1%) | -0.0009 | 537 (98.4%) | 534 (97.8%) | 0.0006 | 1138.67 (0.43) | 1156.05 (0.43) | 0.000 |
| 2019; n (%) | 2,039 (48.0%) | 1,996 (47.0%) | 0.0015 | NA | NA | NA | NA | NA | NA |
| 2020; n (%) | 990 (23.3%) | 1,013 (23.8%) | -0.0010 | NA | NA | NA | NA. | NA | NA |
| Age* | 330 (23.370) | 1,015 (25.070) | 0.0010 | 191 | | | | | |
| mean (sd) | 69.91 (9.75) | 69.94 (9.22) | -0.0032 | 63.70 (10.74) | 63.68 (9.77) | 0.0019 | 69.20 (9.87) | 69.23 (9.28) | -0.003 |
| median [IQR] | 71.00 [64.00, 77.00] | 71.00 [64.00, 76.00] | | 62.00 [57.00, 70.00] | 62.00 [57.00, 70.00] | 0.0000 | 69.97 (9.87) | 69.97 (9.28) | 0.000 |
| Age categories | 7 1.00 (0 1.00, 7 7.00) | 7 1.00 (0 1.00, 7 0.00) | 0.0000 | 02.00 [57.00, 70.00] | 02.00 [57.00, 70.00] | 0.0000 | 03.37 (3.07) | 03.37 (3.20) | 0.000 |
| 40-64; n (%) | 1,154 (27.2%) | 1,129 (26.6%) | 0.0012 | 357 (65.4%) | 364 (66.7%) | -0.0016 | 1,511 (31.5%) | 1,493 (31.1%) | 0.009 |
| 65 - 74; n (%) | 1,682 (39.6%) | 1,714 (40.3%) | -0.0011 | 87 (15.9%) | 87 (15.9%) | 0.0000 | 1,769 (36.9%) | 1,801 (37.6%) | -0.014 |
| | 1,412 (33.2%) | | 0.0001 | 102 (18.7%) | 95 (17.4%) | 0.0031 | 1,514 (31.6%) | 1,500 (31.3%) | 0.006 |
| >= 75; n (%) | 1,412 (33.2/0) | 1,405 (33.1%) | 0.0002 | 102 (10.770) | 33 (17.470) | 0.0031 | 1,514 (51.0%) | 1,300 (31.3%) | 0.000 |
| Geographic Region* | 412 (0.70/) | 404 (0.5%) | 0.0000 | 114/20 00/\ | 112/20 50/\ | 0.0009 | E27/11 00/1 | E16 (10 00/) | 0.000 |
| Northeast; n (%) | 413 (9.7%) | 404 (9.5%) | 0.0006 | 114 (20.9%) | 112 (20.5%) | | 527 (11.0%) | 516 (10.8%) | 0.006 |
| North Central; n (%) | NA 2 444 (57 50() | NA | NA<br>0.0000 | 122 (22.3%) | 121 (22.2%) | 0.0002 | NA 2 722 (5 6 00() | NA | NA |
| South; n (%) | 2,444 (57.5%) | 2,443 (57.5%) | 0.0000 | 278 (50.9%) | 273 (50.0%) | 0.0013 | 2,722 (56.8%) | 2,716 (56.7%) | 0.002 |
| Midwest; n (%) | 776 (18.3%) | 792 (18.6%) | -0.0007 | NA | NA | NA | NA | NA | NA |
| West; n (%) | 615 (14.5%) | 609 (14.3%) | 0.0005 | 32 (5.9%) | 40 (7.3%) | -0.0055 | 647 (13.5%) | 649 (13.5%) | 0.000 |
| Unknown/Missing; n (%) | NA | NA | NA | 0 (0.0%) | 0 (0.0%) | - | NA | NA | NA |
| General Health Related Measures | | | | | | | | | |
| moking; n (%)* | 1,987 (46.8%) | 2,011 (47.3%) | -0.0007 | 254 (46.5%) | 245 (44.9%) | 0.0024 | 2,241 (46.7%) | 2,256 (47.1%) | -0.008 |
| lcohol/Drug abuse or dependence ; n (%) | 264 (6.2%) | 261 (6.1%) | 0.0004 | 21 (3.8%) | 21 (3.8%) | 0.0000 | 285 (5.9%) | 282 (5.9%) | 0.000 |
| Dbesity or Overweight; n (%)* | 1,287 (30.3%) | 1,323 (31.1%) | -0.0014 | 132 (24.2%) | 146 (26.7%) | -0.0050 | 1,419 (29.6%) | 1,469 (30.6%) | -0.022 |
| Dbesity; n (%) | 947 (22.3%) | 945 (22.2%) | 0.0002 | 105 (19.2%) | 117 (21.4%) | -0.0049 | 1,052 (21.9%) | 1,062 (22.2%) | -0.00 |
| Overweight; n (%) | 411 (9.7%) | 456 (10.7%) | -0.0031 | 35 (6.4%) | 36 (6.6%) | -0.0008 | 446 (9.3%) | 492 (10.3%) | -0.034 |
| Cardiovascular Measures | | | | | | | | | |
| Hypertension; n (%)* | 3,229 (76.0%) | 3,262 (76.8%) | -0.0009 | 336 (61.5%) | 342 (62.6%) | -0.0014 | 3,565 (74.4%) | 3,604 (75.2%) | -0.018 |
| Hyperlipidemia; n (%)* | 2,122 (50.0%) | 2,114 (49.8%) | 0.0003 | 203 (37.2%) | 208 (38.1%) | -0.0015 | 2,325 (48.5%) | 2,322 (48.4%) | 0.002 |
| All, angina, Coronary atherosclerosis and other forms of chronic schemic heart disease; n (%)* | 1,047 (24.6%) | 1,043 (24.6%) | 0.0000 | 97 (17.8%) | 106 (19.4%) | -0.0037 | 1,144 (23.9%) | 1,149 (24.0%) | -0.002 |
| Old MI; n (%) | 166 (3.9%) | 155 (3.6%) | 0.0015 | 9 (1.6%) | 5 (0.9%) | 0.0063 | 175 (3.7%) | 160 (3.3%) | 0.022 |
| Acute MI; n (%) | 0 (0.0%) | 0 (0.0%) | 0.0013 | 3 (0.5%) | 0 (0.0%) | 0.0100 | 003 (0.1%) | 000 (0.0%) | 0.022 |
| Stable angina; n (%) | 193 (4.5%) | 187 (4.4%) | 0.0005 | 21 (3.8%) | 23 (4.2%) | -0.0020 | 214 (4.5%) | 210 (4.4%) | 0.045 |
| | 193 (4.3%) | 107 (4.470) | 0.0003 | 21 (5.0%) | 23 (4.2%) | -0.0020 | 214 (4.5%) | 210 (4.4%) | 0.003 |
| Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 971 (22.9%) | 958 (22.6%) | 0.0006 | 89 (16.3%) | 96 (17.6%) | -0.0032 | 1,060 (22.1%) | 1,054 (22.0%) | 0.002 |
| History of CABG or PTCA; n (%) | 268 (6.3%) | 260 (6.1%) | 0.0008 | 12 (2.2%) | 14 (2.6%) | -0.0026 | 280 (5.8%) | 274 (5.7%) | 0.004 |
| Cerebrovascular disease (Stroke, TIA, Late effects); n (%)* | 166 (3.9%) | 169 (4.0%) | -0.0005 | 11 (2.0%) | 15 (2.7%) | -0.0046 | 177 (3.7%) | 184 (3.8%) | -0.005 |
| troke (Ischemic or hemorrhagic); n (%) | 88 (2.1%) | 101 (2.4%) | -0.0020 | 7 (1.3%) | 9 (1.6%) | -0.0025 | 095 (2.0%) | 110 (2.3%) | -0.021 |
| ΠΑ; n (%) | 61 (1.4%) | 58 (1.4%) | 0.0000 | 6 (1.1%) | 6 (1.1%) | 0.0000 | 067 (1.4%) | 064 (1.3%) | 0.009 |
| ate effects of cerebrovascular disease; n (%) | 60 (1.4%) | 59 (1.4%) | 0.0000 | 0 (0.0%) | 2 (0.4%) | -0.0089 | 060 (1.3%) | 061 (1.3%) | 0.000 |
| Atrial fibrillation and Other cardiac dysrhythmia; n (%)* | 707 (16.6%) | 688 (16.2%) | 0.0010 | 67 (12.3%) | 72 (13.2%) | -0.0025 | 774 (16.1%) | 760 (15.9%) | 0.005 |
| Atrial fibrillation; n (%) | 467 (11.0%) | 474 (11.2%) | -0.0006 | 47 (8.6%) | 43 (7.9%) | 0.0024 | 514 (10.7%) | 517 (10.8%) | -0.003 |
| Other cardiac dysrhythmia; n (%) | 707 (16.6%) | 688 (16.2%) | 0.0010 | 67 (12.3%) | 72 (13.2%) | -0.0025 | 774 (16.1%) | 760 (15.9%) | 0.005 |
| Diabetes Related Measures | . , , | (/ | | - 1 1 | | | ,/ | (/ | |
| Diabetes with or w/o complications; n (%)* | 1,151 (27.1%) | 1,149 (27.0%) | 0.0002 | 106 (19.4%) | 110 (20.1%) | -0.0016 | 1,257 (26.2%) | 1,259 (26.3%) | -0.002 |
| Diabetes mellitus without mention of complications; n (%) | 969 (22.8%) | 989 (23.3%) | -0.0010 | 94 (17.2%) | 96 (17.6%) | -0.0010 | 1,063 (22.2%) | 1,085 (22.6%) | -0.010 |
| Diabetes with specified complications; n (%) | 471 (11.1%) | 441 (10.4%) | 0.0010 | 38 (7.0%) | 33 (6.0%) | 0.0039 | 509 (10.6%) | 474 (9.9%) | 0.023 |
| Diabetes with unspecified complications; n (%) | 84 (2.0%) | 102 (2.4%) | -0.0027 | 17 (3.1%) | 7 (1.3%) | 0.0033 | 101 (2.1%) | 109 (2.3%) | -0.014 |
| Gl Conditions | 04 (2.070) | 102 (2.470) | 3.0027 | 17 (3.170) | / (1.3/0) | 0.0121 | 101 (2.170) | 103 (2.3/0) | -0.012 |
| | 1.067 (25.10/) | 1.000 (25.10) | 0.0000 | 0.0 (17.00/) | 100 (10 00/) | 0.0044 | 1 165 (24 20) | 1 176 (24 564) | 0.00 |
| GERD; n (%)* | 1,067 (25.1%) | 1,068 (25.1%) | 0.0000 | 98 (17.9%) | 108 (19.8%) | -0.0044 | 1,165 (24.3%) | 1,176 (24.5%) | -0.00 |
| Jpper GI (Diseases of esophagus, stomach and duodenum including SERD) ; n (%) | 1,149 (27.0%) | 1,166 (27.4%) | -0.0008 | 118 (21.6%) | 117 (21.4%) | 0.0004 | 1,267 (26.4%) | 1,283 (26.8%) | -0.00 |
| Gl bleeding; n (%)* | 100 (2.4%) | 104 (2.4%) | 0.0000 | 14 (2.6%) | 14 (2.6%) | 0.0000 | 114 (2.4%) | 118 (2.5%) | -0.00 |
| Non-infective enteritis and colitis; n (%) | 110 (2.6%) | 103 (2.4%) | 0.0013 | 12 (2.2%) | 13 (2.4%) | -0.0013 | 122 (2.5%) | 116 (2.4%) | 0.00 |

| Intraoperative and postprocedural complications and disorders of | 82 (1.9%) | 73 (1.7%) | 0.0015 | 9 (1.6%) | 9 (1.6%) | 0.0000 | 091 (1.9%) | 082 (1.7%) | 0.015 |
|---|---|---|---|---|---|---|---|---|---|
| digestive system; n (%) | ` ′ | , , | | , , | | | , , | , , | |
| Disorders of gallbladder, biliary tract and pancreas; n (%)* | 92 (2.2%) | 89 (2.1%) | 0.0007 | 11 (2.0%) | 12 (2.2%) | -0.0014 | 103 (2.1%) | 101 (2.1%) | 0.000 |
| Rheumatic Conditions | | | | | | | | | |
| Rheumatoid arthritis and other inflammatory polyarthropathies; n (%)* | 142 (3.3%) | 148 (3.5%) | -0.0011 | 16 (2.9%) | 14 (2.6%) | 0.0018 | 158 (3.3%) | 162 (3.4%) | -0.006 |
| Osteoarthrosis; n (%)* | 1,006 (23.7%) | 1,014 (23.9%) | -0.0004 | 85 (15.6%) | 82 (15.0%) | 0.0015 | 1,091 (22.8%) | 1,096 (22.9%) | -0.002 |
| Other rheumatic disorders (including gout); n (%)* | 1,738 (40.9%) | 1,755 (41.3%) | -0.0006 | 155 (28.4%) | 161 (29.5%) | -0.0020 | 1,893 (39.5%) | 1,916 (40.0%) | -0.010 |
| Gout and other crystal arthropathies; n (%) | 147 (3.5%) | 142 (3.3%) | 0.0011 | 7 (1.3%) | 6 (1.1%) | 0.0018 | 154 (3.2%) | 148 (3.1%) | 0.006 |
| Other rheumatic disorders; n (%) | 1,666 (39.2%) | 1,676 (39.5%) | -0.0005 | 150 (27.5%) | 159 (29.1%) | -0.0030 | 1,816 (37.9%) | 1,835 (38.3%) | -0.008 |
| Neuro Conditions | | | | | | | | | |
| Alzheimer and other Dementia Disease ; n (%)* | 191 (4.5%) | 185 (4.4%) | 0.0005 | 8 (1.5%) | 7 (1.3%) | 0.0017 | 199 (4.2%) | 192 (4.0%) | 0.010 |
| Seizure disorders (epilepsy); n (%)* | 69 (1.6%) | 64 (1.5%) | 0.0008 | 0 (0.0%) | 2 (0.4%) | -0.0089 | 069 (1.4%) | 066 (1.4%) | 0.000 |
| Delirium/Psychosis; n (%)* | 118 (2.8%) | 116 (2.7%) | 0.0006 | 9 (1.6%) | 5 (0.9%) | 0.0063 | 127 (2.6%) | 121 (2.5%) | 0.006 |
| Other Conditions | | | | | | | | | |
| Hypothyroidism; n (%)* | 748 (17.6%) | 744 (17.5%) | 0.0002 | 84 (15.4%) | 76 (13.9%) | 0.0039 | 832 (17.4%) | 820 (17.1%) | 0.008 |
| Chronic kidney disease stages I-III; n (%)* | 646 (15.2%) | 663 (15.6%) | -0.0010 | 31 (5.7%) | 33 (6.0%) | -0.0012 | 677 (14.1%) | 696 (14.5%) | -0.011 |
| Chronic kidney disease stages IV-V, ESRD; n (%) | 87 (2.0%) | 86 (2.0%) | 0.0000 | 7 (1.3%) | 4 (0.7%) | 0.0060 | 094 (2.0%) | 090 (1.9%) | 0.007 |
| COPD; n (%) | 3,860 (90.9%) | 4,087 (96.2%) | -0.0055 | 503 (92.1%) | 527 (96.5%) | -0.0046 | 4,363 (91.0%) | 4,614 (96.2%) | -0.214 |
| Asthma; n (%)* | 988 (23.3%) | 1,018 (24.0%) | -0.0014 | 149 (27.3%) | 140 (25.6%) | 0.0033 | 1,137 (23.7%) | 1,158 (24.2%) | -0.012 |
| Obstructive sleep apnea; n (%)* | 870 (20.5%) | 890 (21.0%) | -0.0011 | 104 (19.0%) | 118 (21.6%) | -0.0058 | 974 (20.3%) | 1,008 (21.0%) | -0.017 |
| Syncope; n (%) | 134 (3.2%) | 120 (2.8%) | 0.0023 | 14 (2.6%) | 9 (1.6%) | 0.0069 | 148 (3.1%) | 129 (2.7%) | 0.024 |
| Falls; n (%) | 227 (5.3%) | 237 (5.6%) | -0.0013 | 10 (1.8%) | 12 (2.2%) | -0.0028 | 237 (4.9%) | 249 (5.2%) | -0.014 |
| VTE; n (%)* | 119 (2.8%) | 121 (2.8%) | 0.0000 | 9 (1.6%) | 8 (1.5%) | 0.0008 | 128 (2.7%) | 129 (2.7%) | 0.000 |
| Combined comorbidity score, 365 days* | | | | | | | | | |
| mean (sd) | 3.14 (2.58) | 3.14 (2.63) | 0.0000 | 2.22 (2.09) | 2.27 (2.07) | -0.0240 | 3.04 (2.53) | 3.04 (2.57) | 0.000 |
| median [IQR] | 3.00 [1.00, 5.00] | 2.00 [1.00, 5.00] | 0.3839 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.0000 | 2.89 (2.53) | 2.00 (2.57) | 0.349 |
| INDEX 2 - Frailty Score: Empirical Version 365 days as Categories, | 3.00 [1.00, 3.00] | 2.00 [1.00, 5.00] | 0.3633 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.0000 | 2.89 (2.55) | 2.00 (2.57) | 0.343 |
| v3* | | | | | | | | | |
| <0.1 non frail; n (%) | 3,304 (77.8%) | 3,296 (77.6%) | 0.0002 | 417 (76.4%) | 418 (76.6%) | -0.0002 | 3,721 (77.6%) | 3,714 (77.5%) | 0.002 |
| 0.1 -<0.2 prefrail; n (%) | 786 (18.5%) | 801 (18.9%) | -0.0009 | 111 (20.3%) | 108 (19.8%) | 0.0011 | 897 (18.7%) | 909 (19.0%) | -0.008 |
| > 0.2 frail; n (%) | 158 (3.7%) | 151 (3.6%) | 0.0005 | 18 (3.3%) | 20 (3.7%) | -0.0021 | 176 (3.7%) | 171 (3.6%) | 0.005 |
| Medication Use | , , | , , | | , , | , , | | . , | , , | |
| Use of oral corticosteroids; n (%)* | 3,931 (92.5%) | 3,936 (92.7%) | -0.0002 | 528 (96.7%) | 522 (95.6%) | 0.0011 | 4,459 (93.0%) | 4,458 (93.0%) | 0.000 |
| Use of antidepressants; n (%)* | 1,804 (42.5%) | 1,817 (42.8%) | -0.0005 | 226 (41.4%) | 221 (40.5%) | 0.0014 | 2,030 (42.3%) | 2,038 (42.5%) | -0.004 |
| Use of anticonvulsants; n (%)* | 1,070 (25.2%) | 1,083 (25.5%) | -0.0006 | 97 (17.8%) | 97 (17.8%) | 0.0000 | 1,167 (24.3%) | 1,180 (24.6%) | -0.007 |
| Use of beta blocker OR calcium channel blocker; n (%)* | 1,672 (39.4%) | 1,679 (39.5%) | -0.0002 | 177 (32.4%) | 174 (31.9%) | 0.0009 | 1,849 (38.6%) | 1,853 (38.7%) | -0.002 |
| Use of PPIs; n (%)* | 1,461 (34.4%) | 1,498 (35.3%) | -0.0015 | 174 (31.9%) | 178 (32.6%) | -0.0012 | 1,635 (34.1%) | 1,676 (35.0%) | -0.019 |
| Use of opioids; n (%)* | 1,358 (32.0%) | 1,360 (32.0%) | 0.0000 | 149 (27.3%) | 150 (27.5%) | -0.0004 | 1,507 (31.4%) | 1,510 (31.5%) | -0.002 |
| Use of antipsychotics; n (%)* | 221 (5.2%) | 222 (5.2%) | 0.0000 | 25 (4.6%) | 25 (4.6%) | 0.0000 | 246 (5.1%) | 247 (5.2%) | -0.005 |
| Use of anxiolytics/hypnotics; n (%)* | 416 (9.8%) | 420 (9.9%) | -0.0003 | 55 (10.1%) | 56 (10.3%) | -0.0006 | 471 (9.8%) | 476 (9.9%) | -0.003 |
| Use of dementia meds; n (%)* | 122 (2.9%) | 134 (3.2%) | -0.0017 | 5 (0.9%) | 4 (0.7%) | 0.0022 | 127 (2.6%) | 138 (2.9%) | -0.018 |
| Use of antiparkinsonian meds; n (%)* | 204 (4.8%) | 194 (4.6%) | 0.0009 | 22 (4.0%) | 18 (3.3%) | 0.0037 | 226 (4.7%) | 212 (4.4%) | 0.014 |
| Use of Benzodiazepine; n (%)* | 850 (20.0%) | 854 (20.1%) | -0.0002 | 111 (20.3%) | 110 (20.1%) | 0.0004 | 961 (20.0%) | 964 (20.1%) | -0.002 |
| All antidiabetic medications; n (%)* | 901 (21.2%) | 907 (21.4%) | -0.0004 | 99 (18.1%) | 107 (19.6%) | -0.0035 | 1,000 (20.9%) | 1,014 (21.2%) | -0.007 |
| ACEI/ARB; n (%)* | 2,013 (47.4%) | 2,018 (47.5%) | -0.0001 | 225 (41.2%) | 231 (42.3%) | -0.0017 | 2,238 (46.7%) | 2,249 (46.9%) | -0.004 |
| Use of Anticoagulants; n (%)* | 446 (10.5%) | 449 (10.6%) | -0.0003 | 48 (8.8%) | 50 (9.2%) | -0.0013 | 494 (10.3%) | 499 (10.4%) | -0.003 |
| Use of Amiodarone; n (%) | 46 (1.1%) | 54 (1.3%) | -0.0018 | 4 (0.7%) | 6 (1.1%) | -0.0042 | 050 (1.0%) | 060 (1.3%) | -0.028 |
| Digoxin; n (%) | 51 (1.2%) | 51 (1.2%) | 0.0000 | 3 (0.5%) | 6 (1.1%) | -0.0067 | 054 (1.1%) | 057 (1.2%) | -0.009 |
| Use of Diuretics; n (%)* | 1,653 (38.9%) | 1,668 (39.3%) | -0.0006 | 193 (35.3%) | 192 (35.2%) | 0.0002 | 1,846 (38.5%) | 1,860 (38.8%) | -0.006 |
| Use of Aspirin; n (%) | 19 (0.4%) | 30 (0.7%) | -0.0040 | 12 (2.2%) | 12 (2.2%) | 0.0000 | 031 (0.6%) | 042 (0.9%) | -0.035 |
| NSAIDs (NOT including aspirin); n (%) | 742 (17.5%) | 741 (17.4%) | 0.0002 | 112 (20.5%) | 95 (17.4%) | 0.0071 | 854 (17.8%) | 836 (17.4%) | 0.011 |
| HRT (Use of estrogens, progestins, androgens); n (%)* | 142 (3.3%) | 142 (3.3%) | 0.0000 | 28 (5.1%) | 36 (6.6%) | -0.0062 | 170 (3.5%) | 178 (3.7%) | -0.011 |
| Use of Statins ; n (%)* | 2,335 (55.0%) | 2,355 (55.4%) | -0.0005 | 244 (44.7%) | 234 (42.9%) | 0.0027 | 2,579 (53.8%) | 2,589 (54.0%) | -0.004 |
| Healthcare Utilization Measures | | | | | | | | | |
| Use of any drugs claims* | | | | | | | | | |
| mean (sd) | 38.70 (25.02) | 38.49 (22.66) | 0.0088 | 38.41 (24.47) | 38.81 (22.54) | -0.0170 | 38.67 (24.96) | 38.53 (22.65) | 0.006 |
| median [IQR] | 34.00 [21.00, 51.00] | 34.00 [22.00, 50.00 | 0.0000 | 34.50 [21.00, 50.25] | 35.00 [23.00, 50.00] | -0.0213 | 34.06 (24.96) | 34.11 (22.65) | -0.002 |
| Number of office visits* | 18.87 (12.67) | 18.79 (12.49) | 0.0064 | 14.24 (9.91) | 14.60 (9.82) | -0.0365 | 18.34 (12.39) | | 0.002 |

| | _ | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| median [IQR] | 16.00 [10.00, 24.75] | 16.00 [10.00, 24.00] | 0.0000 | 12.00 [7.00, 18.00] | 12.00 [8.00, 19.00] | 0.0000 | 15.54 (12.39) | 15.54 (12.22) | 0.000 |
| Number of ED visits* | | | | | | | | | |
| mean (sd) | 1.19 (1.76) | 1.19 (1.95) | 0.0000 | 0.99 (1.47) | 1.02 (1.70) | -0.0189 | 1.17 (1.73) | 1.17 (1.92) | 0.000 |
| median [IQR] | 1.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | 0.0000 | 0.00 [0.00, 1.00] | 0.00 [0.00, 2.00] | 0.0000 | 0.89 (1.73) | 0.89 (1.92) | 0.000 |
| Number of hospitalizations* | | | | | | | | | |
| mean (sd) | 0.17 (0.52) | 0.18 (0.57) | -0.0183 | 0.89 (2.85) | 0.86 (2.33) | 0.0115 | 0.25 (1.08) | 0.26 (0.95) | -0.010 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (1.08) | 0.00 (0.95) | 0.000 |
| Recent hospitalization (-30 days to Index Rx date); n (%)* | 71 (1.7%) | 66 (1.6%) | 0.0008 | 8 (1.5%) | 6 (1.1%) | 0.0035 | 079 (1.6%) | 072 (1.5%) | 0.008 |
| Old hospitalizations (-365 to -31 days); n (%)* | 1,070 (25.2%) | 1,098 (25.8%) | -0.0012 | 144 (26.4%) | 146 (26.7%) | -0.0006 | 1,214 (25.3%) | 1,244 (25.9%) | -0.014 |
| Number of Pulmonologist visits* | | | | | | | | | |
| mean (sd) | 0.09 (0.67) | 0.09 (0.61) | 0.0000 | 1.08 (1.76) | 1.15 (1.49) | -0.0429 | 0.20 (0.87) | 0.21 (0.76) | -0.012 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 2.00] | 1.00 [0.00, 2.00] | -0.6133 | 0.00 (0.87) | 0.11 (0.76) | -0.135 |
| Pulmonologist on CED ; n (%)* | 24 (0.6%) | 23 (0.5%) | 0.0013 | 55 (10.1%) | 61 (11.2%) | -0.0034 | 079 (1.6%) | 084 (1.8%) | -0.015 |
| Number of hospital days* | | | | | | | | | |
| mean (sd) | 1.25 (5.14) | 1.29 (6.09) | -0.0071 | 0.89 (2.85) | 0.86 (2.33) | 0.0115 | 1.21 (4.93) | 1.24 (5.79) | -0.006 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.0000 | 0.00 (4.93) | 0.00 (5.79) | 0.000 |
| Occurrence of basic or comprehensive metabolic blood chemistry | 2.000/00.00/\ | 2,903 (68.3%) | -0.0004 | 256 (46.9%) | 252 (46. 20/) | 0.0010 | 2 144 (CE CO/) | 2 155 (65 80/) | -0.004 |
| test; n (%)* | 2,888 (68.0%) | 2,903 (08.3%) | -0.0004 | 250 (40.9%) | 252 (46.2%) | 0.0010 | 3,144 (65.6%) | 3,155 (65.8%) | -0.004 |
| Number of HbA1C test ordered* | | | | | | | | | |
| mean (sd) | 1.11 (1.45) | 1.11 (1.46) | 0.0000 | 0.58 (1.08) | 0.61 (1.18) | -0.0265 | 1.05 (1.41) | 1.05 (1.43) | 0.000 |
| median [IQR] | 1.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.6873 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.0000 | 0.89 (1.41) | 0.00 (1.43) | 0.627 |
| Flexible Sigmoidoscopy or colonoscopy or CT virtual colonoscopy; | 171 (4.0%) | 169 (4.0%) | 0.0000 | 27 (4.9%) | 32 (5.9%) | -0.0043 | 198 (4.1%) | 201 (4.2%) | -0.005 |
| n (%)* | 171 (4.0%) | 109 (4.0%) | 0.0000 | 27 (4.5%) | 32 (3.3%) | -0.0043 | 190 (4.1%) | 201 (4.2%) | -0.003 |
| Number of Mammograms (Breast cancer screening); n (%)* | 534 (12.6%) | 529 (12.5%) | 0.0003 | 62 (11.4%) | 64 (11.7%) | -0.0009 | 596 (12.4%) | 593 (12.4%) | 0.000 |
| Number of Pap smear (Cervical cancer screening); n (%)* | 86 (2.0%) | 97 (2.3%) | -0.0020 | 18 (3.3%) | 20 (3.7%) | -0.0021 | 104 (2.2%) | 117 (2.4%) | -0.013 |
| Flu vaccine; n (%)* | 865 (20.4%) | 852 (20.1%) | 0.0007 | 85 (15.6%) | 90 (16.5%) | -0.0022 | 950 (19.8%) | 942 (19.6%) | 0.005 |
| Pneumococcal vaccine; n (%)* | 1,184 (27.9%) | 1,149 (27.0%) | 0.0017 | 107 (19.6%) | 114 (20.9%) | -0.0029 | 1,291 (26.9%) | 1,263 (26.3%) | 0.014 |
| Copay for pharmacy cost (charges in U.S. \$)* | | | | | | | | | |
| mean (sd) | 27.30 (35.49) | 27.85 (31.85) | -0.0163 | 21.53 (22.71) | 20.69 (20.10) | 0.0392 | 26.64 (34.28) | 27.03 (30.74) | -0.012 |
| median [IQR] | 19.37 [6.01, 36.26] | 20.58 [6.59, 38.83] | -0.0359 | 16.99 [7.47, 28.40] | 17.25 [9.01, 26.47] | -0.0121 | 19.10 (34.28) | 20.20 (30.74) | -0.034 |
| SES 9 Proxy - Business Type* | | | | | | | | | |
| Commercial; n (%) | 605 (14.2%) | 586 (13.8%) | 0.0011 | NA | NA | NA | NA | NA | NA |
| Medicare; n (%) | 3,643 (85.8%) | 3,662 (86.2%) | -0.0004 | NA | NA | NA | NA | NA | NA |
| SABA Copy; n (%)* | 2,502 (58.9%) | 2,495 (58.7%) | 0.0003 | 387 (70.9%) | 377 (69.0%) | 0.0023 | 2,889 (60.3%) | 2,872 (59.9%) | 0.008 |
| SAMA; n (%)* | 176 (4.1%) | 189 (4.4%) | -0.0015 | 32 (5.9%) | 28 (5.1%) | 0.0034 | 208 (4.3%) | 217 (4.5%) | -0.010 |
| SABA/SAMA Copy; n (%)* | 757 (17.8%) | 763 (18.0%) | -0.0005 | 113 (20.7%) | 105 (19.2%) | 0.0034 | 870 (18.1%) | 868 (18.1%) | 0.000 |
| ICS Copy; n (%)* | 856 (20.2%) | 870 (20.5%) | -0.0007 | 142 (26.0%) | 150 (27.5%) | -0.0029 | 998 (20.8%) | 1,020 (21.3%) | -0.012 |
| LABA Copy; n (%)* | 37 (0.9%) | 40 (0.9%) | 0.0000 | 5 (0.9%) | 8 (1.5%) | -0.0055 | 042 (0.9%) | 048 (1.0%) | -0.010 |
| LAMA Copy; n (%)* | 918 (21.6%) | 926 (21.8%) | -0.0004 | 189 (34.6%) | 177 (32.4%) | 0.0038 | 1,107 (23.1%) | 1,103 (23.0%) | 0.002 |
| LABA/ICS Combination Copy; n (%) | 4,248 (100.0%) | 1,462 (34.4%) | 0.0804 | 546 (100.0%) | 254 (46.5%) | 0.0628 | 4,794 (100.0%) | 1,716 (35.8%) | 1.894 |
| LAMA/LABA Combination Copy; n (%)* | 301 (7.1%) | 312 (7.3%) | -0.0007 | 65 (11.9%) | 73 (13.4%) | -0.0042 | 366 (7.6%) | 385 (8.0%) | -0.015 |
| LABA LAMA ICS Copy; n (%) | 0 (0.0%) | 4,248 (100.0%) | -0.1421 | 0 (0.0%) | 546 (100.0%) | -0.1421 | 000 (0.0%) | 4,794 (100.0%) | - |
| GOLD C/D status; n (%)* | 3,022 (71.1%) | 3,021 (71.1%) | 0.0000 | 387 (70.9%) | 378 (69.2%) | 0.0020 | 3,409 (71.1%) | 3,399 (70.9%) | 0.004 |
| blood eosinophilia test; n (%)* | 14 (0.3%) | 15 (0.4%) | -0.0017 | 3 (0.5%) | 3 (0.5%) | 0.0000 | 017 (0.4%) | 018 (0.4%) | 0.000 |
| Serum immunoglobulin E (IgE) level test Copy; n (%)* | 100 (2.4%) | 94 (2.2%) | 0.0013 | 13 (2.4%) | 15 (2.7%) | -0.0019 | 113 (2.4%) | 109 (2.3%) | 0.007 |
| H2 blocker; n (%)* | 340 (8.0%) | 336 (7.9%) | 0.0004 | 30 (5.5%) | 31 (5.7%) | -0.0008 | 370 (7.7%) | 367 (7.7%) | 0.000 |
| Oxygen codes; n (%)* | 396 (9.3%) | 413 (9.7%) | -0.0013 | 61 (11.2%) | 61 (11.2%) | 0.0000 | 457 (9.5%) | 474 (9.9%) | -0.014 |
| Respiratory arrest/dependence on oxygen; n (%)* | 501 (11.8%) | 516 (12.1%) | -0.0009 | 70 (12.8%) | 69 (12.6%) | 0.0006 | 571 (11.9%) | 585 (12.2%) | -0.009 |
| Insurance Plan Type* | 1 | | | | | | | | |
| Comprehensive; n (%) | Ī | NA | NA | 63 (11.5%) | 68 (12.5%) | -0.0029 | NA | NA | NA |
| comprenensive, ir (70) | NA | | | | 55 (10.1%) | -0.0006 | NA | NA | NA |
| HMO; n (%) | NA<br>NA | NA | NA | 54 (9.9%) | 55 (10.1%) | -0.0000 | INA | INA | |
| | | | NA<br>NA | 54 (9.9%)<br>287 (52.6%) | 289 (52.9%) | -0.0004 | NA | NA | NA |
| HMO; n (%) | NA | NA | | | | | | | NA<br>NA |
| HMO; n (%)<br>PPO; n (%) | NA<br>NA | NA<br>NA | NA | 287 (52.6%) | 289 (52.9%) | -0.0004 | NA | NA | |
| HMO; n (%)<br>PPO; n (%)<br>Others; n (%) | NA<br>NA | NA<br>NA | NA | 287 (52.6%) | 289 (52.9%) | -0.0004<br>0.0030<br>0.0021 | NA | NA | |
| HMO; n (%)PPO; n (%)Others; n (%) Metropolitan Statistical Area* | NA<br>NA<br>NA | NA<br>NA<br>NA | NA<br>NA | 287 (52.6%)<br>142 (26.0%) | 289 (52.9%)<br>134 (24.5%) | -0.0004<br>0.0030 | NA<br>NA | NA<br>NA | NA |

<sup>\*</sup>Included in the 1:1 PS matching model